Replication of the D58 Asthma Trial in Healthcare Claims Data

**DUPLICATE-D58** 

September 14, 2021

NCT04892732

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

A 26 Week, Randomized, Double-blind, Parallel-group, Active Controlled, Multicenter, Multinational Safety Study Evaluating the Risk of Serious Asthma-related Events During Treatment With Symbicort®, a Fixed Combination of Inhaled Corticosteroid (ICS) (Budesonide) and a Long Acting β2-agonist (LABA) (Formoterol) as Compared to Treatment With ICS (Budesonide) Alone in Adult and Adolescent (≥12 Years of Age) Patients With Asthma (D5896C00027 Study NCT01444430)

#### 1.2 Intended aim(s)

To assess the effects of 26 weeks treatment with budesonide-formoterol compared with budesonide alone on the incidence of first serious asthma-related event (a composite of adjudicated death, intubation, and hospitalization) in patients who had persistent asthma.

# 1.3 Primary endpoint for replication

First serious asthma-related event (a composite of adjudicated death, intubation, and hospitalization.

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

To meet the prespecified noninferiority margin, the upper limit of the two-sided 95% confidence interval of the hazard ratio for the first serious asthma-related event with budesonide-formoterol versus budesonide had to be less than 2.0. The incidence rate of serious asthma-related events in the budesonide-only treatment group was predicted to be 0.0075 over a 26-week period. It was calculated that 87 events would have to occur for the study to have 90% power to rule out an event rate with budesonide-formoterol that was twice as high as the rate with budesonide alone.

# 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Individual components of the primary outcome 1) Asthma-related hospitalization

- 2) Asthma-related intubation
- 3) Asthma-related death

#### 1.6 Trial estimate

Hazard Ratio, HR = 1.07 (95% CI, 0.70 to 1.65) comparing budesonide-formoterol versus budesonide during a 26-week period (Peters et al., 2016).

# 2. Person responsible for implementation of replication in Aetion

Hemin Lee, MD, MPH, implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum CDM, IBM® MarketScan®

# 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1. Design Diagram - D5896C00027 (NCT 01444430) TRIAL REPLICATION



#### 5. Cohort Identification

### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing budesonide-formoterol versus budesonide alone. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of budesonide-formoterol or budesonide.

### 5.2 Important steps for cohort formation

New use of budesonide-formoterol (exposure) is defined as no use of the exposure drug within the 180 days prior to index date. This will emulate the trial requirement for which treatment with budesonide-formoterol was not allowed any time before randomization. New use of budesonide (comparator) is defined as no use of the comparator drug within the 180 days prior to index date. New users of budesonide are not allowed to receive of budesonide-formoterol within the 180 days prior to index date, and new users of budesonide-formoterol are not allowed to receive budesonide within the 180 days prior to index date.

### 5.2.1 Eligible cohort entry dates

Budesonide-formoterol was approved by FDA on July 21, 2006 for management of asthma. The initial eligible cohort entry date was the first date after July 21, 2006 for both the databases investigated (IBM® MarketScan®, Optum CDM). The last date eligible as cohort entry date was the end of available data for IBM® MarketScan® and Optum CDM. The following eligible cohort entry dates were included:

- IBM® MarketScan®: July 21, 2006 December 31, 2018 (end of available data)
- Optum CDM: July 21, 2006 June 30, 2020 (end of available data)
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

# 5.3 Flowchart of the study cohort assembly For Budesonide-formoterol vs. Budesonide

| | Optun | n CDM | IBM® MarketScan® | |
|---|---|---|---|---|
| Less Excluded Patients | Remaining<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78,202,636 | | 200,203,908 |
| Did not meet cohort entry criteria | -<br>77,464,646 | 737,990 | -<br>198,996,061 | 1,207,847 |
| Excluded due to insufficient enrollment | -114,685 | 623,305 | -157,484 | 1,050,363 |
| Excluded due to prior use of referent | -27,092 | 596,213 | -80,459 | 969,904 |
| Excluded due to prior use of exposure | -292,949 | 303,264 | -398,899 | 571,005 |
| Excluded because patient qualified in >1 exposure category | -40 | 303,224 | -139 | 570,866 |
| Excluded based on Age: exclude missing | -3 | 303,221 | 0 | 570,866 |
| Excluded based on Gender: exclude missing | 0 | 303,221 | 0 | 570,866 |
| Excluded based on INCLUSION: Age >=12 | -14,027 | 289,194 | -38,285 | 532,581 |
| Excluded based on Inclusion 2 - Asthma >=1 year prior to CED | -167,426 | 121,768 | -316,772 | 215,809 |
| Excluded based on Inclusion 3 - Asthma exacerbation (combination) [-365,-30] | -59,930 | 61,838 | -150,606 | 65,203 |
| Excluded based on Inclusion 4 - Asthma Therapy [-365,-30] | -10,146 | 51,692 | -8,560 | 56,643 |
| Excluded based on Exclusion 1 - Acute respiratory failure - intubation/nivs (combination) | -4,103 | 47,589 | -3,423 | 53,220 |
| Excluded based on Exclusion 2b - Asthma exacerbation (combination) >4 in 365 days | -5,195 | 42,394 | -3,857 | 49,363 |
| Excluded based on Exclusion 2C - Asthma exacerbation (inpatient primary) >2 times in 365 days | -4,020 | 38,374 | -109 | 49,254 |
| Excluded based on Exclusion 3 - Use of oral corticosteroids (-30, 0] | -3,222 | 35,152 | -6,184 | 43,070 |
| Excluded based on Exclusion 4 - Asthma exacerbation (combination) [-7,0] | -196 | 34,956 | -483 | 42,587 |
| Excluded based on Exclusion 7 - Respiratory disease (combination) | -540 | 34,416 | -609 | 41,978 |
| Excluded based on Exclusion 8 - Smoking | -931 | 33,485 | -657 | 41,321 |
| Excluded based on Exclusion 9 - Acute upper or lower respiratory infections | -2,527 | 30,958 | -4,278 | 37,043 |
| Excluded based on Exclusion 10 - Pregnancy | -66 | 30,892 | -85 | 36,958 |
| Excluded based on Exclusion 11 - Malignancy | -308 | 30,584 | -367 | 36,591 |
| Excluded based on Exclusion 14 - Use of omalizumab | -1 | 30,583 | -103 | 36,488 |

| Excluded based on Exclusion 15 - Use of Beta-blocker | -150 | 30,433 | -161 | 36,327 |
|---|---|---|---|---|
| Excluded based on Exclusion 19 - Drug/alcohol abuse | -49 | 30,384 | -31 | 36,296 |
| Final cohort | | 30,384 | | 36,296 |

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

New initiation of Budesonide-formoterol (80/4.5 ug or 160/4.5 ug twice daily). New initiation is defined as no use of Budesonide-formoterol in the prior **180** days before treatment initiation (washout period). New users of Budesonide-formoterol are not allowed to receive budesonide within the 180 days prior to treatment initiation.

#### Comparator agent:

New initiation of Budesonide alone. New initiation is defined as no use of budesonide in the prior 180 days before treatment initiation (washout period). New users of budesonide are not allowed to receive Budesonide-formoterol within the 180 days prior to treatment initiation.

# 6.2 <u>Preliminary Covariates:</u>

- Age
- Gender
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date.

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**).

# 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- **Primary outcome**: First serious asthma-related event (a composite of adjudicated death, intubation, and hospitalization **Secondary outcome**: Individual components of the primary outcome 1) Asthma-related hospitalization
  - 2) Asthma-related intubation
  - 3) Asthma-related death

# 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the primary analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of Budesonide-formoterol and Budesonide and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continuous registration in the database,
- Discontinuation of the index drugs,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (Budesonide-formoterol or a comparator) plus a defined grace period (i.e., 60 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation
  - A dosage change on the index treatment does not fulfill this criterion

## 7. Initial Feasibility Analysis

Action report name:

#### For Budesonide-formoterol vs. budesonide

Optum CDM - https://bwh-dope.aetion.com/projects/details/1657/results/67114/result/0

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1656/results/67113/result/0

Date conducted: 03/16/2021

Complete Aetion feasibility analysis using age and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

#### 8. Initial Power Assessment

#### Aetion report name:

- For Budesonide-formoterol vs. budesonide
- Optum CDM https://bwh-dope.aetion.com/projects/details/1657/rwrs/67089
   IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1656/rwrs/67108

Date conducted: 03/17/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, gender, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 3/19/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 4/2/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

For Budesonide-formoterol vs. budesonide

Optum CDM: https://bwh-dope.aetion.com/projects/details/1657/rwrs/68456 IBM® MarketScan®: https://bwh-dope.aetion.com/projects/details/1656/rwrs/68455

Date conducted: 4/14/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

- Provide plot of PS distributions stratified by treatment group. Note- Please refer to **Appendix B**.
- Report covariate balance after matching.

  Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 14 (0.06%) | 5 (0.02%) | 9 (0.04%) |
| Start of an additional exposure | 291 (1.20%) | 242 (1.00%) | 49 (0.20%) |
| End of index exposure | 20257 (83.31%) | 10172 (41.84%) | 10085 (41.48%) |
| Specified date reached | 486 (2.00%) | 227 (0.93%) | 259 (1.07%) |
| End of patient data | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| End of patient enrollment | 3159 (12.99%) | 1463 (6.02%) | 1696 (6.98%) |
| Nursing home admission, pharmacy disenrollment | 107 (0.44%) | 48 (0.20%) | 59 (0.24%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|------------------------------------|--------------|---------------|
| Patient Group | Optum | Marketscan |
| Overall Patient Population | 88 [88,148] | 107 [88,163] |
| Referent – | 88 [88,148] | 93 [88, 148] |
| Exposure | 88 [88, 158] | 116 [88, 177] |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | Pooled |
|-------------------------|-----------|------------------|--------|
| Risk per 1,000 patients | 3.7 | 4.7 | 4.2 |

# 10. Final Power Assessment

Date conducted: 4/15/2021

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.
  - o <u>Pooled</u>

| Non-inferiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 24,314 |
| Reference | 12,157 |
| Exposed | 12,157 |
| Risk per 1,000 patients | 4.2 |
| Assumed HR from RCT | 1.07 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 102.1188 |
| Power | 0.885015194 |

o Optum CDM

| Optum CDM | |
|----------------------------|-------------|
| Non-inferiority Analysis | |
| Number of patients matched | 10,396 |
| Reference | 5,198 |
| Exposed | 5,198 |
| Risk per 1,000 patients | 3.7 |
| Assumed HR from RCT | 1.07 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 38.4652 |
| Power | 0.491896419 |

o IBM® MarketScan®

| Non-inferiority Analysis | |
|----------------------------|------------|
| Number of patients matched | 13,918 |
| Reference | 6,959 |
| Exposed | 6,959 |
| Risk per 1,000 patients | 4.7 |
| Assumed HR from RCT | 1.07 |
| Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 2 |
| Number of events expected | 65.4146 |
| Power | 0.71548801 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 4/16/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 4/30/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

# 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u> Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the

individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

# 12. Register study protocol on clinicalTrials.gov

### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

# 13. Comparative Analyses

Action report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 <u>For sensitivity analyses:</u>

# 14. Requested Results

# 14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

# 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

# 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

# 14.5 <u>Table 5: Results from secondary analyses.</u>

# 15. References

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177.

| | | | | Color Coding Criteria |
|---|---|---|---|---|
| # | NCT01444430 trial definitions | Implementation in routine care | Please see the following Google Drive for further details or any missing information:<br>https://drive.google.com/drive/folders/1WD618wrywYjEaXzfl.TcuK-VCcnb6b-gV?usp=sharing | Can be replicated in claims |
| | | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive | Using dummy definitions for measuring in claims |
| | | | Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/ backward mapping based on the CMS ICD-9 to ICD-10 | Can't be measured in claims |
| | | | mapping:<br>https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk-general-equivalence- | |
| | Trial details- clinicaltrial.gov NCT0144443 EXPOSURE vs. COMPARISON | 8 | Reference/Rationale | Can't be measured in claims but not important for the analysis |
| | Exposure) Budesonide-formoterol<br>Referent) Budesonide | Exposure: Budesonide-formoterol Two actuations of 80 ug of budesonide plus 4.5 ug of formoterol or 160 ug of budesonide plus 4.5 ug of formoterol) NDC code: 0186037020 - budesonide/formoterol fumarate 00186037020 - budesonide/formoterol fumarate 00186037220 - budesonide/formoterol fumarate 00186037220 - budesonide/formoterol fumarate 00186037220 - budesonide/formoterol fumarate 54569646600 - budesonide/formoterol fumarate 54569646600 - budesonide/formoterol fumarate 54686593700 - budesonide/formoterol fumarate 84686593700 - budesonide/formoterol fumarate 84686593700 - budesonide/formoterol fumarate 86686593700 - budesonide/formoterol fumarate 8676964600 - budesonide/formoterol fumarate 86769700 - budesonide/formoterol fumarate 87700 - budesonide/formoterol fumarate 87800 - budesonide/formoterol fumarate 87800 - budesonide/formoterol fumarate 87800 - budesonide/formoterol fumarate 88800 - budesonide/formoterol fumarate 88800 - budesonide/formoterol fumarate 88800 - budesonide/formoterol fumarate 88800 - budesonide/formoterol fumarate 98800 - budesonide/formoterol fumarate 988000 - budesonide/formoterol fumarate 988000 - budesonide/formoterol fumarate 988000 - budesonide/ | | |
| 1 | PRIMARY OUTCOME | | | |
| | First Serious asthma-related events<br>(Composite of asthma-related deaths, intubations, and hospitalizations) | Measured 1 day after drug initiationo in inpatient setting Asthma-related death: Inpatient death with primary discharge code of asthma (Optum, Marketscan) + Patient attribute for death (Optum) Asthma related -Intubations: Diagnosis code for asthma in primary position plus CPT procedure code, 31500: Endotracheal intubation, emergency in inpatient or Emergency room setting Asthma-related Hospitalizations: Inpatient discharge diagnosis for asthma in primary position | | |
| | INCLUSION CRITERIA | | | |
| 1 | | Measured on the day of drug initiation | | |
| 1 | INCLUSION CRITERIA 212 years of age | Measured on the day of drug initiation Age >= 12 | | |
| | | | Larsson K, Ställberg B, Lisspers K, Telg G, Johansson G, Thuresson M, Janson C. Prevalence and management of severe asthma in primary care: an observational cohort study in Sweden (PACEHR), Respir Res. 2018 Jan 18;19(1):12. doi: 10.1186/s12931-018-0719-x PMID: 29347939; PMID: PMC5774144. | |
| 2 | ≥12 years of age | $Age>=12$ Measured between [- $\infty$ , 365] days prior to drug initiation in any position/any setting Asthma: ICD-9:493x | management of severe asthma in primary care: an observational cohort study in Sweden (PACEHR). Respir Res. 2018 Jan 18;19(1):12. doi: 10.1186/s12931-018-0719-x. PMID: | |
| 3 | 212 years of age Documented clinical diagnosis of asthma for ≥1 year prior to randomization History of at least one asthma exacerbation in the previous year (but none in the 4 weeks prior to randomization. An asthma exacerbation was defined as an event requiring treatment with systemic corticosteroids or requiring hospitalization (i.e. an inpatient stay or >24-hour stay in | Age >= 12 Measured between [-∞, 365] days prior to drug initiation in any position/any setting Asthma: ICD-9. 493x ICD-10: 145.* Measured between 30 to 365 days prior to drug initiation in defined position and setting 1) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code Asthma: ICD-9. 493x | management of severe asthma in primary care: an observational cohort study in Sweden (PACEHR). Respir Res. 2018 Jan 18;19(1):12. doi: 10.1186/s12931-018-0719-x. PMID: | |
| 3 | Documented clinical diagnosis of asthma for 21 year prior to randomization History of at least one authma exacerbation in the previous year (but none in the 4 weeks prior to randomization. An asthma exacerbation was defined as an event requiring treatment with systemic conticosteroids or requiring hospitalization (i.e. an inpatient stay or >24-hour stay in the observation area of an emergency room or local equivalent) | Age >= 12 Measured between [-0, 365] days prior to drug initiation in any position/any setting Asthma: ICD-9: 493x ICD-10: 145.* Measured between 30 to 365 days prior to drug initiation in defined position and setting 1) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code Asthma: ICD-9: 493x ICD-10: 145.* Measured between 30 to 365 days prior to drug initiation in defined position and setting Aprescription claim for one of the following asthma maintenance medications: ICS monotherapy ICS/LABA combination: Xanthines Leukotriene receptor antagonist | management of severe asthma in primary care: an observational cohort study in Sweden (PACEHR). Respir Res. 2018 Jan 18;19(1):12. doi: 10.1186/s12931-018-0719-x. PMID: | |
| 3 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | Documented clinical diagnosis of asthma for 21 year prior to randomization History of at least one asthma exacerbation in the previous year (but none in the 4 weeks prior to randomization. An asthma exacerbation was defined as an event requiring treatment with systemic corticosteroids or requiring hospitalization (i.e. an inpatient stay or >24-hour stay in the observation area of an emergency room or local equivalent) Receiving: A stable dose of ICS alone or in combination with a LABA, leukotriene receptor antagonist or other maintenance therapy/therapies for 24 weeks prior to randomization (any patient maintained on a stable high-dose ICS with or without a LABA or LTRA or other maintenance therapy/therapies was required to have an ACQ6 total score of <1.5 at screening) or | Age >= 12 Measured between [-∞, 365] days prior to drug initiation in any position/any setting Asthma: ICD-0.493x ICD-0.1945.* Measured between 30 to 365 days prior to drug initiation in defined position and setting 1) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code Asthma: ICD-0.9493x ICD-10: 45.* Measured between 30 to 365 days prior to drug initiation in defined position and setting Measured between 30 to 365 days prior to drug initiation in defined position and setting ICS/LABA combination: Xanthines Leukotriene receptor antagonist Note) Did not incorporate SABA as it is difficult to capture daily use | management of severe asthma in primary care: an observational cohort study in Sweden (PACEHR). Respir Res. 2018 Jan 18;19(1):12. doi: 10.1186/s12931-018-0719-x. PMID: | |
| 3 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | Documented clinical diagnosis of asthma for ≥1 year prior to randomization History of at least one asthma exacerbation in the previous year (but none in the 4 weeks prior to randomization. An asthma exacerbation was defined as an event requiring treatment with systemic corticosteroids or requiring hospitalization (i.e. an inpatient stay or >24-hour stay in the observation area of an emergency room or local equivalent) Receiving: A stable dose of ICS alone or in combination with a LABA, leukotriene receptor antagonist or other maintenance therapy/therapies for ≥4 weeks prior to randomization (any patient maintained on a stable high-dose ICS with or without a LABA or LTRA or other maintenance therapy/therapies was required to have an ACQ6 total score of <1.5 at screening) or A stable dose of LTRA or xanthine monotherapy (for ≥4 weeks prior to randomization) or daily SABA (in the 4 weeks before randomization but \$8 puffs a day on two consecutive days, or ≥25 puffs in one day, in the 7 days prior to screening. | Age >= 12 Measured between [-0, 365] days prior to drug initiation in any position/any setting Asthma: ICD-9: 493x ICD-10: 145.* Measured between 30 to 365 days prior to drug initiation in defined position and setting 1) Asthma diagnosis code in inpatient primary diagnosis position 2) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code Asthma: ICD-9: 493x ICD-10: 145.* Measured between 30 to 365 days prior to drug initiation in defined position and setting Aprescription claim for one of the following asthma maintenance medications: ICS monotherapy ICS/LABA combination: Xanthines Leukotriene receptor antagonist | management of severe asthma in primary care: an observational cohort study in Sweden (PACEHR). Respir Res. 2018 Jan 18;19(1):12. doi: 10.1186/s12931-018-0719-x. PMID: | |

Color Coding Criteria

| | Measured any time prior to and including drug initiation date in any setting | Walkey AJ, Wiener RS. Use of noninvasive ventilation in patients with acute respiratory failure, |
|---|---|---|
| A history of life-threatening asthma (defined as an asthma episode that required intubation and/or was associated with hypercapnia requiring non-invasive ventilatory support) | Acute respiratory failure/insufficiency/arrest (EO-9:513-7;518.2",518.8",518.8",518.83", "518.84", "799.1", "V46.1", "V46.11", "V46.12", "V46.13", "V46.21" (EO-10:-190", "196.00", "196.01", "196.02", "196.11", "196.12", "196.20", "196.21", "196.22", "196.00", "196.11", "196.92", "809.01", "809.2", "729.11", "729.12", "299.81") Intubation/Non-invasive ventilatory support: (EO-9 Procedure code: "93.90", "93.92", "96.01", "96.02", "96.03", "96.04", "96.05", "96.70", "96.71", "96.72" (EO-10 procedure codes: "09.1018.22", "09.118.22", "08.112.22", "08.112.22", "08.113.22", " | 2000-2009: a population-based study. Ann Am Thorac Soc. 2013 Feb;10(1):10-7. doi: 10.1513/AnnalsATS.201206-0340C. PMID: 23509327; PMCID: PMC3780971. |
| 2a) Any asthma exacerbation requiring systemic corticosteroids within 4 weeks prior to randomization or 2(b)>4 separate exacerbations or 2(c)>2 separate exacerbations or 2(c)>2 hospitalizations (an inpatient stay or >24-hour stay in the observation area of an emergency room or local equivalent) due to asthma in the previous year | 2c) Asthma hospitalization, measured >2 times, 365 days prior to drug initiation Asthma: ICD-9:493.x ICD-10:145.* | http://mchp-appserv.cpe.umanitoba.ca/concept/asthma_table1.html |
| 3 Received systemic corticosteroids for any reason in the 4 weeks prior to randomization | Measured 30 days prior to and including the day of drug initiation Cortisone, hydrocortisone, prednisone, prednisolone, methylprednisolone, triamcinolone, dexamethasone, betamethasone | |
| 4 Had an ongoing asthma exacerbation requiring systemic corticosteroids | Measured 7 days prior to aind including the day of drug initiation Asthma exacerbation Defined as a) Asthma diagnosis code in inpatient primary diagnosis position b) Asthma diagnosis code in inpatient any position or outpatient setting PLUS a prescription claim for systemic steroids 14 days before and after the diagnosis code Asthma: ICD-9: 493.x ICD-10: 145.* | |
| Unstable asthma within 7 days prior to randomization (defined as asthma symptoms that persisted throughout the day on two consecutive days, night-time awakening due to asthma during 23 nights, rescue medication use for the acute worsening of asthma symptoms of x8 inhalations aday over two consecutive days or 225 inhalations in one day, and asthma symptoms so severe that the patient was limited in their ability to perform normal daily activity) | N/A | |
| 6 Peak expiratory flow (pre- or post-bronchodilatory) <50% of predicted normal | N/A | |
| Concurrent respiratory disease (chronic obstructive pulmonary disease, chronic bronchitis, emphysema, idiopathic pulmonary fibrosis, bronchiectasis, and/or any pulmonary disease) | Secastre 180 days prior to drug mination in any care setting and position | |
| 8 A smoking history of >10 pack-years | V15.82, 305.1x, 649.0x, 989.84 OR CPT code 99406, 99407, G0436, G0437, G9016, S9075, S9453, S4995, G9276, G9458, 1034F, 4004F, 4001F OR UNITED THE CONTROL OF THE CONTROL | |
| 9 Respiratory infection or other viral/bacterial illness | Measured 180 days prior to drug initiation in any position/any setting Acute upper /lower respiratory infections ICD-10: 00.x 01.x 02.x 03.x 04.x 05.x 06.x 20.x 21.x 22.x | |
| 10 Pregnancy (current/planned) and lactation | Measured 180 days prior to drug initiation in any position/any setting See tab [Pregnancy] | |
| | | · |

| 11 | Malignancy (with the exception of basal cell carcinoma) within the 5 years prior to study commencement | Measured 180 days prior to drug initiation in any position/any setting |
|---|---|---|
| 11 | mangnancy (with the exception of basal central minutes) within the 5 years prior to study commencement | See tab [Malignancy] |
| 12 | Known or suspected hypersensitivity to study medications or their excipients | N/A |
| 13 | Participation in a concurrent LABA safety study or other interventional or investigational drug study | N/A |
| 1/1 | Omalizumab or any other monoclonal/polyclonal antibody use in the 6 months prior to randomization | Measured 180 days prior to drug initiation |
| 14 | Omanzamas or any other monocional porycional antibody usem the omorths prior to randomization | Drug generic name: omalizumab |
| | | Measured 30 days prior to drug initiation |
| 15 | Concomitant β-blocker use | Druggeneric name: Propranolo, bucindolol, carteolol, carvedilol, labetalol, nadolol, Oxprenolol, penbutolol, pindolol, sotalol, timolol, Acebutolol, Atenolol, Betaxolol, bisoprolol, Celiprolol, metoprolol, nebivolol, esmolol, butaxamine, nebivolol |
| 16 | Any other significant disease/disorder that, in the opinion of the investigator, could have either put the patient at risk, or influence the results of the study or the patient's ability to participate in the study | N/A |
| 17 | Clinically relevant abnormal findings in physical examination/vital signs at randomization | N/A |
| 18 | Risk of non-compliance | N/A |
| 19 | Drug/alcohol abuse | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care settling. Alcohol abuse or dependence: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drugabuse or dependence: 292.xx, 304.xx, 305.2x-305.9x, 648.3x |
| 20 | Planned blood donation during the study | N/A |
| 21 | Affiliation with study sponsor and/or investigator | N/A |

# Pregnancy Diagnosis codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN+A2:J81 V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY Procedure codes 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION 72.4 FORCEPS ROTATION OF FETAL HEAD 72.5 BREECH EXTRACTION

72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD

72.52 OTHER PARTIAL BREECH EXTRACTION

- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
  72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION
- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

#### Malignancy 140 - MALIGNANT NEOPLASM OF LIP 140.0 - MALIGNANT NEOPLASM OF UPPER LIP VERMILION BORDER 140.1 - MALIGNANT NEOPLASM OF LOWER LIP VERMILION BORDER 140.3 - MALIGNANT NEOPLASM OF UPPER LIP INNER ASPECT 140.4 - MALIGNANT NEOPLASM OF LOWER LIP INNER ASPECT 140.5 - MALIGNANT NEOPLASM OF LIP UNSPECIFIED INNER ASPECT 140.6 - MALIGNANT NEOPLASM OF COMMISSURE OF LIP 140.8 - MALIGNANT NEOPLASM OF OTHER SITES OF LIP 140.9 - MALIGNANT NEOPLASM OF LIP UNSPECIFIED VERMILION BORDER 141 - MALIGNANT NEOPLASM OF TONGUE 141.0 - MALIGNANT NEOPLASM OF BASE OF TONGUE 141.1 - MALIGNANT NEOPLASM OF DORSAL SURFACE OF TONGUE 141.2 - MALIGNANT NEOPLASM OF TIP AND LATERAL BORDER OF TONGUE 141.3 - MALIGNANT NEOPLASM OF VENTRAL SURFACE OF TONGUE 141.4 - MALIGNANT NEOPLASM OF ANTERIOR TWO-THIRDS OF TONGUE PART UNSPECIFIED 141.5 - MALIGNANT NEOPLASM OF JUNCTIONAL ZONE OF TONGUE 141.6 - MALIGNANT NEOPLASM OF LINGUAL TONSIL 141.8 - MALIGNANT NEOPLASM OF OTHER SITES OF TONGUE 141.9 - MALIGNANT NEOPLASM OF TONGUE UNSPECIFIED 142 - MALIGNANT NEOPLASM OF MAJOR SALIVARY GLANDS 142.0 - MALIGNANT NEOPLASM OF PAROTID GLAND 142.1 - MALIGNANT NEOPLASM OF SUBMANDIBULAR GLAND 142.2 - MALIGNANT NEOPLASM OF SUBLINGUAL GLAND 142.8 - MALIGNANT NEOPLASM OF OTHER MAJOR SALIVARY GLANDS 142.9 - MALIGNANT NEOPLASM OF SALIVARY GLAND UNSPECIFIED 143 - MALIGNANT NEOPLASM OF GUM 143.0 - MALIGNANT NEOPLASM OF UPPER GUM 143.1 - MALIGNANT NEOPLASM OF LOWER GUM 143.8 - MALIGNANT NEOPLASM OF OTHER SITES OF GUM 143.9 - MALIGNANT NEOPLASM OF GUM UNSPECIFIED 144 - MALIGNANT NEOPLASM OF FLOOR OF MOUTH 144.0 - MALIGNANT NEOPLASM OF ANTERIOR PORTION OF FLOOR OF MOUTH 144.1 - MALIGNANT NEOPLASM OF LATERAL PORTION OF FLOOR OF MOUTH 144.8 - MALIGNANT NEOPLASM OF OTHER SITES OF FLOOR OF MOUTH 144.9 - MALIGNANT NEOPLASM OF FLOOR OF MOUTH PART UNSPECIFIED 145 - MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF MOUTH 145.0 - MALIGNANT NEOPLASM OF CHEEK MUCOSA 145.1 - MALIGNANT NEOPLASM OF VESTIBULE OF MOUTH 145.2 - MALIGNANT NEOPLASM OF HARD PALATE 145.3 - MALIGNANT NEOPLASM OF SOFT PALATE 145.4 - MALIGNANT NEOPLASM OF UVULA 145.5 - MALIGNANT NEOPLASM OF PALATE UNSPECIFIED 145.6 - MALIGNANT NEOPLASM OF RETROMOLAR AREA 145.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED PARTS OF MOUTH 145.9 - MALIGNANT NEOPLASM OF MOUTH UNSPECIFIED

- 146 MALIGNANT NEOPLASM OF OROPHARYNX 146.0 - MALIGNANT NEOPLASM OF TONSIL 146.1 - MALIGNANT NEOPLASM OF TONSILLAR FOSSA 146.2 - MALIGNANT NEOPLASM OF TONSILLAR PILLARS (ANTERIOR) (POSTERIOR) 146.3 - MALIGNANT NEOPLASM OF VALLECULA EPIGLOTTICA 146.4 - MALIGNANT NEOPLASM OF ANTERIOR ASPECT OF EPIGLOTTIS 146.5 - MALIGNANT NEOPLASM OF JUNCTIONAL REGION OF OROPHARYNX 146.6 - MALIGNANT NEOPLASM OF LATERAL WALL OF OROPHARYNX 146.7 - MALIGNANT NEOPLASM OF POSTERIOR WALL OF OROPHARYNX 146.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF OROPHARYNX 146.9 - MALIGNANT NEOPLASM OF OROPHARYNX UNSPECIFIED SITE 147 - MALIGNANT NEOPLASM OF NASOPHARYNX 147.0 - MALIGNANT NEOPLASM OF SUPERIOR WALL OF NASOPHARYNX 147.1 - MALIGNANT NEOPLASM OF POSTERIOR WALL OF NASOPHARYNX 147.2 - MALIGNANT NEOPLASM OF LATERAL WALL OF NASOPHARYNX 147.3 - MALIGNANT NEOPLASM OF ANTERIOR WALL OF NASOPHARYNX 147.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF NASOPHARYNX 147.9 - MALIGNANT NEOPLASM OF NASOPHARYNX UNSPECIFIED SITE 148 - MALIGNANT NEOPLASM OF HYPOPHARYNX 148.0 - MALIGNANT NEOPLASM OF POSTCRICOID REGION OF HYPOPHARYNX 148.1 - MALIGNANT NEOPLASM OF PYRIFORM SINUS 148.2 - MALIGNANT NEOPLASM OF ARYEPIGLOTTIC FOLD HYPOPHARYNGEAL ASPECT 148.3 - MALIGNANT NEOPLASM OF POSTERIOR HYPOPHARYNGEAL WALL 148.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF HYPOPHARYNX 148.9 - MALIGNANT NEOPLASM OF HYPOPHARYNX UNSPECIFIED SITE 149 - MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES WITHIN THE LIP ORAL CAVITY AND PHARYNX 149.0 - MALIGNANT NEOPLASM OF PHARYNX UNSPECIFIED 149.1 - MALIGNANT NEOPLASM OF WALDEYER'S RING 149.8 - MALIGNANT NEOPLASM OF OTHER SITES WITHIN THE LIP AND ORAL CAVITY 149.9 - MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITHIN THE LIP AND ORAL CAVITY 150 - MALIGNANT NEOPLASM OF ESOPHAGUS 150.0 - MALIGNANT NEOPLASM OF CERVICAL ESOPHAGUS 150.1 - MALIGNANT NEOPLASM OF THORACIC ESOPHAGUS 150.2 - MALIGNANT NEOPLASM OF ABDOMINAL ESOPHAGUS 150.3 - MALIGNANT NEOPLASM OF UPPER THIRD OF ESOPHAGUS 150.4 - MALIGNANT NEOPLASM OF MIDDLE THIRD OF ESOPHAGUS 150.5 - MALIGNANT NEOPLASM OF LOWER THIRD OF ESOPHAGUS 150.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED PART OF ESOPHAGUS 150.9 - MALIGNANT NEOPLASM OF ESOPHAGUS UNSPECIFIED SITE 151 - MALIGNANT NEOPLASM OF STOMACH 151.0 - MALIGNANT NEOPLASM OF CARDIA 151.1 - MALIGNANT NEOPLASM OF PYLORUS 151.2 - MALIGNANT NEOPLASM OF PYLORIC ANTRUM
- 151.4 MALIGNANT NEOPLASM OF BODY OF STOMACH 151.5 - MALIGNANT NEOPLASM OF LESSER CURVATURE OF STOMACH UNSPECIFIED

151.3 - MALIGNANT NEOPLASM OF FUNDUS OF STOMACH

- 151.6 MALIGNANT NEOPLASM OF GREATER CURVATURE OF STOMACH UNSPECIFIED
- 151.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF STOMACH
- 151.9 MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED SITE
- 152 MALIGNANT NEOPLASM OF SMALL INTESTINE INCLUDING DUODENUM
- 152.0 MALIGNANT NEOPLASM OF DUODENUM
- 152.1 MALIGNANT NEOPLASM OF JEJUNUM
- 152.2 MALIGNANT NEOPLASM OF ILEUM
- 152.3 MALIGNANT NEOPLASM OF MECKEL'S DIVERTICULUM
- 152.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF SMALL INTESTINE
- 152.9 MALIGNANT NEOPLASM OF SMALL INTESTINE UNSPECIFIED SITE
- 153 MALIGNANT NEOPLASM OF COLON
- 153.0 MALIGNANT NEOPLASM OF HEPATIC FLEXURE
- 153.1 MALIGNANT NEOPLASM OF TRANSVERSE COLON
- 153.2 MALIGNANT NEOPLASM OF DESCENDING COLON
- 153.3 MALIGNANT NEOPLASM OF SIGMOID COLON
- 153.4 MALIGNANT NEOPLASM OF CECUM
- 153.5 MALIGNANT NEOPLASM OF APPENDIX VERMIFORMIS
- 153.6 MALIGNANT NEOPLASM OF ASCENDING COLON
- 153.7 MALIGNANT NEOPLASM OF SPLENIC FLEXURE
- 153.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF LARGE INTESTINE
- 153.9 MALIGNANT NEOPLASM OF COLON UNSPECIFIED SITE
- 154 MALIGNANT NEOPLASM OF RECTUM RECTOSIGMOID JUNCTION AND ANUS
- 154.0 MALIGNANT NEOPLASM OF RECTOSIGMOID JUNCTION
- 154.1 MALIGNANT NEOPLASM OF RECTUM
- 154.2 MALIGNANT NEOPLASM OF ANAL CANAL
- 154.3 MALIGNANT NEOPLASM OF ANUS UNSPECIFIED SITE
- 154.8 MALIGNANT NEOPLASM OF OTHER SITES OF RECTUM RECTOSIGMOID JUNCTION AND ANUS
- 155 MALIGNANT NEOPLASM OF LIVER AND INTRAHEPATIC BILE DUCTS
- 155.0 MALIGNANT NEOPLASM OF LIVER PRIMARY
- 155.1 MALIGNANT NEOPLASM OF INTRAHEPATIC BILE DUCTS
- 155.2 MALIGNANT NEOPLASM OF LIVER NOT SPECIFIED AS PRIMARY OR SECONDARY
- 156 MALIGNANT NEOPLASM OF GALLBLADDER AND EXTRAHEPATIC BILE DUCTS
- 156.0 MALIGNANT NEOPLASM OF GALLBLADDER
- 156.1 MALIGNANT NEOPLASM OF EXTRAHEPATIC BILE DUCTS
- 156.2 MALIGNANT NEOPLASM OF AMPULLA OF VATER
- 156.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF GALLBLADDER AND EXTRAHEPATIC BILE DUCTS
- 156.9 MALIGNANT NEOPLASM OF BILIARY TRACT PART UNSPECIFIED SITE
- 157 MALIGNANT NEOPLASM OF PANCREAS
- 157.0 MALIGNANT NEOPLASM OF HEAD OF PANCREAS
- 157.1 MALIGNANT NEOPLASM OF BODY OF PANCREAS
- 157.2 MALIGNANT NEOPLASM OF TAIL OF PANCREAS
- 157.3 MALIGNANT NEOPLASM OF PANCREATIC DUCT
- 157.4 MALIGNANT NEOPLASM OF ISLETS OF LANGERHANS
- 157.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF PANCREAS
- 157.9 MALIGNANT NEOPLASM OF PANCREAS PART UNSPECIFIED
- 158 MALIGNANT NEOPLASM OF RETROPERITONEUM AND PERITONEUM

- 158.0 MALIGNANT NEOPLASM OF RETROPERITONEUM
- 158.8 MALIGNANT NEOPLASM OF SPECIFIED PARTS OF PERITONEUM
- 158.9 MALIGNANT NEOPLASM OF PERITONEUM UNSPECIFIED
- 159 MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES WITHIN THE DIGESTIVE ORGANS AND PERITONEUM
- 159.0 MALIGNANT NEOPLASM OF INTESTINAL TRACT PART UNSPECIFIED
- 159.1 MALIGNANT NEOPLASM OF SPLEEN NOT ELSEWHERE CLASSIFIED
- 159.8 MALIGNANT NEOPLASM OF OTHER SITES OF DIGESTIVE SYSTEM AND INTRA-ABDOMINAL ORGANS
- 159.9 MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITHIN THE DIGESTIVE ORGANS AND PERITONEUM
- 160 MALIGNANT NEOPLASM OF NASAL CAVITIES MIDDLE EAR AND ACCESSORY SINUSES
- 160.0 MALIGNANT NEOPLASM OF NASAL CAVITIES
- 160.1 MALIGNANT NEOPLASM OF AUDITORY TUBE MIDDLE EAR AND MASTOID AIR CELLS
- 160.2 MALIGNANT NEOPLASM OF MAXILLARY SINUS
- 160.3 MALIGNANT NEOPLASM OF ETHMOIDAL SINUS
- 160.4 MALIGNANT NEOPLASM OF FRONTAL SINUS
- 160.5 MALIGNANT NEOPLASM OF SPHENOIDAL SINUS
- 160.8 MALIGNANT NEOPLASM OF OTHER ACCESSORY SINUSES
- 160.9 MALIGNANT NEOPLASM OF ACCESSORY SINUS UNSPECIFIED
- 161 MALIGNANT NEOPLASM OF LARYNX
- 161.0 MALIGNANT NEOPLASM OF GLOTTIS
- 161.1 MALIGNANT NEOPLASM OF SUPRAGLOTTIS
- 161.2 MALIGNANT NEOPLASM OF SUBGLOTTIS
- 161.3 MALIGNANT NEOPLASM OF LARYNGEAL CARTILAGES
- 161.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF LARYNX
- 161.9 MALIGNANT NEOPLASM OF LARYNX UNSPECIFIED
- 162 MALIGNANT NEOPLASM OF TRACHEA BRONCHUS AND LUNG
- 162.0 MALIGNANT NEOPLASM OF TRACHEA
- 162.2 MALIGNANT NEOPLASM OF MAIN BRONCHUS
- 162.3 MALIGNANT NEOPLASM OF UPPER LOBE BRONCHUS OR LUNG
- 162.4 MALIGNANT NEOPLASM OF MIDDLE LOBE BRONCHUS OR LUNG
- 162.5 MALIGNANT NEOPLASM OF LOWER LOBE BRONCHUS OR LUNG
- 162.8 MALIGNANT NEOPLASM OF OTHER PARTS OF BRONCHUS OR LUNG
- 162.9 MALIGNANT NEOPLASM OF BRONCHUS AND LUNG UNSPECIFIED
- 163 MALIGNANT NEOPLASM OF PLEURA
- 163.0 MALIGNANT NEOPLASM OF PARIETAL PLEURA
- 163.1 MALIGNANT NEOPLASM OF VISCERAL PLEURA
- 163.8 MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF PLEURA
- 163.9 MALIGNANT NEOPLASM OF PLEURA UNSPECIFIED
- 164 MALIGNANT NEOPLASM OF THYMUS HEART AND MEDIASTINUM
- 164.0 MALIGNANT NEOPLASM OF THYMUS
- 164.1 MALIGNANT NEOPLASM OF HEART
- 164.2 MALIGNANT NEOPLASM OF ANTERIOR MEDIASTINUM
- 164.3 MALIGNANT NEOPLASM OF POSTERIOR MEDIASTINUM
- 164.8 MALIGNANT NEOPLASM OF OTHER PARTS OF MEDIASTINUM
- 164.9 MALIGNANT NEOPLASM OF MEDIASTINUM PART UNSPECIFIED
- 165 MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES WITHIN THE RESPIRATORY SYSTEM AND INTRATHORACIC ORGANS
- 165.0 MALIGNANT NEOPLASM OF UPPER RESPIRATORY TRACT PART UNSPECIFIED

165.8 - MALIGNANT NEOPLASM OF OTHER SITES WITHIN THE RESPIRATORY SYSTEM AND INTRATHORACIC ORGANS 165.9 - MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITHIN THE RESPIRATORY SYSTEM 170 - MALIGNANT NEOPLASM OF BONE AND ARTICULAR CARTILAGE 170.0 - MALIGNANT NEOPLASM OF BONES OF SKULL AND FACE EXCEPT MANDIBLE 170.1 - MALIGNANT NEOPLASM OF MANDIBLE 170.2 - MALIGNANT NEOPLASM OF VERTEBRAL COLUMN EXCLUDING SACRUM AND COCCYX 170.3 - MALIGNANT NEOPLASM OF RIBS STERNUM AND CLAVICLE 170.4 - MALIGNANT NEOPLASM OF SCAPULA AND LONG BONES OF UPPER LIMB 170.5 - MALIGNANT NEOPLASM OF SHORT BONES OF UPPER LIMB 170.6 - MALIGNANT NEOPLASM OF PELVIC BONES SACRUM AND COCCYX 170.7 - MALIGNANT NEOPLASM OF LONG BONES OF LOWER LIMB 170.8 - MALIGNANT NEOPLASM OF SHORT BONES OF LOWER LIMB 170.9 - MALIGNANT NEOPLASM OF BONE AND ARTICULAR CARTILAGE SITE UNSPECIFIED 171 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE 171.0 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF HEAD FACE AND NECK 171.2 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF UPPER LIMB INCLUDING SHOULDER 171.3 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF LOWER LIMB INCLUDING HIP 171.4 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF THORAX 171.5 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF ABDOMEN 171.6 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF PELVIS 171.7 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE OF TRUNK UNSPECIFIED 171.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF CONNECTIVE AND OTHER SOFT TISSUE 171.9 - MALIGNANT NEOPLASM OF CONNECTIVE AND OTHER SOFT TISSUE SITE UNSPECIFIED 172 - MALIGNANT MELANOMA OF SKIN 172.0 - MALIGNANT MELANOMA OF SKIN OF LIP 172.1 - MALIGNANT MELANOMA OF SKIN OF EYELID INCLUDING CANTHUS 172.2 - MALIGNANT MELANOMA OF SKIN OF EAR AND EXTERNAL AUDITORY CANAL 172.3 - MALIGNANT MELANOMA OF SKIN OF OTHER AND UNSPECIFIED PARTS OF FACE 172.4 - MALIGNANT MELANOMA OF SKIN OF SCALP AND NECK 172.5 - MALIGNANT MELANOMA OF SKIN OF TRUNK EXCEPT SCROTUM 172.6 - MALIGNANT MELANOMA OF SKIN OF UPPER LIMB INCLUDING SHOULDER 172.7 - MALIGNANT MELANOMA OF SKIN OF LOWER LIMB INCLUDING HIP 172.8 - MALIGNANT MELANOMA OF OTHER SPECIFIED SITES OF SKIN 172.9 - MELANOMA OF SKIN SITE UNSPECIFIED 174 - MALIGNANT NEOPLASM OF FEMALE BREAST 174.0 - MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF FEMALE BREAST 174.1 - MALIGNANT NEOPLASM OF CENTRAL PORTION OF FEMALE BREAST 174.2 - MALIGNANT NEOPLASM OF UPPER-INNER QUADRANT OF FEMALE BREAST 174.3 - MALIGNANT NEOPLASM OF LOWER-INNER QUADRANT OF FEMALE BREAST 174.4 - MALIGNANT NEOPLASM OF UPPER-OUTER QUADRANT OF FEMALE BREAST 174.5 - MALIGNANT NEOPLASM OF LOWER-OUTER QUADRANT OF FEMALE BREAST 174.6 - MALIGNANT NEOPLASM OF AXILLARY TAIL OF FEMALE BREAST 174.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF FEMALE BREAST

174.9 - MALIGNANT NEOPLASM OF BREAST (FEMALE) UNSPECIFIED SITE

175.0 - MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF MALE BREAST

175 - MALIGNANT NEOPLASM OF MALE BREAST

175.9 - MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED SITES OF MALE BREAST 176 - KAPOSI'S SARCOMA 176.0 - KAPOSI'S SARCOMA SKIN 176.1 - KAPOSI'S SARCOMA SOFT TISSUE 176.2 - KAPOSI'S SARCOMA PALATE 176.3 - KAPOSI'S SARCOMA GASTROINTESTINAL SITES 176.4 - KAPOSI'S SARCOMA LUNG 176.5 - KAPOSI'S SARCOMA LYMPH NODES 176.8 - KAPOSI'S SARCOMA OTHER SPECIFIED SITES 176.9 - KAPOSI'S SARCOMA UNSPECIFIED SITE 179 - MALIGNANT NEOPLASM OF UTERUS-PART UNS 180 - MALIGNANT NEOPLASM OF CERVIX UTERI 180.0 - MALIGNANT NEOPLASM OF ENDOCERVIX 180.1 - MALIGNANT NEOPLASM OF EXOCERVIX 180.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF CERVIX 180.9 - MALIGNANT NEOPLASM OF CERVIX UTERI UNSPECIFIED SITE 181 - MALIGNANT NEOPLASM OF PLACENTA 182 - MALIGNANT NEOPLASM OF BODY OF UTERUS 182.0 - MALIGNANT NEOPLASM OF CORPUS UTERI EXCEPT ISTHMUS 182.1 - MALIGNANT NEOPLASM OF ISTHMUS 182.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF BODY OF UTERUS 183 - MALIGNANT NEOPLASM OF OVARY AND OTHER UTERINE ADNEXA 183.0 - MALIGNANT NEOPLASM OF OVARY 183.2 - MALIGNANT NEOPLASM OF FALLOPIAN TUBE 183.3 - MALIGNANT NEOPLASM OF BROAD LIGAMENT OF UTERUS 183.4 - MALIGNANT NEOPLASM OF PARAMETRIUM 183.5 - MALIGNANT NEOPLASM OF ROUND LIGAMENT OF UTERUS 183.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF UTERINE ADNEXA 183.9 - MALIGNANT NEOPLASM OF UTERINE ADNEXA UNSPECIFIED SITE 184 - MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED FEMALE GENITAL ORGANS 184.0 - MALIGNANT NEOPLASM OF VAGINA 184.1 - MALIGNANT NEOPLASM OF LABIA MAJORA 184.2 - MALIGNANT NEOPLASM OF LABIA MINORA 184.3 - MALIGNANT NEOPLASM OF CLITORIS 184.4 - MALIGNANT NEOPLASM OF VULVA UNSPECIFIED SITE 184.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF FEMALE GENITAL ORGANS 184.9 - MALIGNANT NEOPLASM OF FEMALE GENITAL ORGAN SITE UNSPECIFIED 185 - MALIGNANT NEOPLASM OF PROSTATE 186 - MALIGNANT NEOPLASM OF TESTIS 186.0 - MALIGNANT NEOPLASM OF UNDESCENDED TESTIS 186.9 - MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED TESTIS 187 - MALIGNANT NEOPLASM OF PENIS AND OTHER MALE GENITAL ORGANS 187.1 - MALIGNANT NEOPLASM OF PREPUCE 187.2 - MALIGNANT NEOPLASM OF GLANS PENIS 187.3 - MALIGNANT NEOPLASM OF BODY OF PENIS 187.4 - MALIGNANT NEOPLASM OF PENIS PART UNSPECIFIED

187.5 - MALIGNANT NEOPLASM OF EPIDIDYMIS 187.6 - MALIGNANT NEOPLASM OF SPERMATIC CORD 187.7 - MALIGNANT NEOPLASM OF SCROTUM 187.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF MALE GENITAL ORGANS 187.9 - MALIGNANT NEOPLASM OF MALE GENITAL ORGAN SITE UNSPECIFIED 188 - MALIGNANT NEOPLASM OF BLADDER 188.0 - MALIGNANT NEOPLASM OF TRIGONE OF URINARY BLADDER 188.1 - MALIGNANT NEOPLASM OF DOME OF URINARY BLADDER 188.2 - MALIGNANT NEOPLASM OF LATERAL WALL OF URINARY BLADDER 188.3 - MALIGNANT NEOPLASM OF ANTERIOR WALL OF URINARY BLADDER 188.4 - MALIGNANT NEOPLASM OF POSTERIOR WALL OF URINARY BLADDER 188.5 - MALIGNANT NEOPLASM OF BLADDER NECK 188.6 - MALIGNANT NEOPLASM OF URETERIC ORIFICE 188.7 - MALIGNANT NEOPLASM OF URACHUS 188.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF BLADDER 188.9 - MALIGNANT NEOPLASM OF BLADDER PART UNSPECIFIED 189 - MALIGNANT NEOPLASM OF KIDNEY AND OTHER AND UNSPECIFIED URINARY ORGANS 189.0 - MALIGNANT NEOPLASM OF KIDNEY EXCEPT PELVIS 189.1 - MALIGNANT NEOPLASM OF RENAL PELVIS 189.2 - MALIGNANT NEOPLASM OF URETER 189.3 - MALIGNANT NEOPLASM OF URETHRA 189.4 - MALIGNANT NEOPLASM OF PARAURETHRAL GLANDS 189.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF URINARY ORGANS 189.9 - MALIGNANT NEOPLASM OF URINARY ORGAN SITE UNSPECIFIED 190 - MALIGNANT NEOPLASM OF EYE 190.0 - MALIGNANT NEOPLASM OF EYEBALL EXCEPT CONJUNCTIVA CORNEA RETINA AND CHOROID 190.1 - MALIGNANT NEOPLASM OF ORBIT 190.2 - MALIGNANT NEOPLASM OF LACRIMAL GLAND 190.3 - MALIGNANT NEOPLASM OF CONJUNCTIVA 190.4 - MALIGNANT NEOPLASM OF CORNEA 190.5 - MALIGNANT NEOPLASM OF RETINA 190.6 - MALIGNANT NEOPLASM OF CHOROID 190.7 - MALIGNANT NEOPLASM OF LACRIMAL DUCT 190.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF EYE 190.9 - MALIGNANT NEOPLASM OF EYE PART UNSPECIFIED 191 - MALIGNANT NEOPLASM OF BRAIN 191.0 - MALIGNANT NEOPLASM OF CEREBRUM EXCEPT LOBES AND VENTRICLES 191.1 - MALIGNANT NEOPLASM OF FRONTAL LOBE 191.2 - MALIGNANT NEOPLASM OF TEMPORAL LOBE 191.3 - MALIGNANT NEOPLASM OF PARIETAL LOBE 191.4 - MALIGNANT NEOPLASM OF OCCIPITAL LOBE 191.5 - MALIGNANT NEOPLASM OF VENTRICLES 191.6 - MALIGNANT NEOPLASM OF CEREBELLUM NOT OTHERWISE SPECIFIED

191.7 - MALIGNANT NEOPLASM OF BRAIN STEM

191.8 - MALIGNANT NEOPLASM OF OTHER PARTS OF BRAIN 191.9 - MALIGNANT NEOPLASM OF BRAIN UNSPECIFIED SITE

192 - MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF NERVOUS SYSTEM 192.0 - MALIGNANT NEOPLASM OF CRANIAL NERVES 192.1 - MALIGNANT NEOPLASM OF CEREBRAL MENINGES 192.2 - MALIGNANT NEOPLASM OF SPINAL CORD 192.3 - MALIGNANT NEOPLASM OF SPINAL MENINGES 192.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF NERVOUS SYSTEM 192.9 - MALIGNANT NEOPLASM OF NERVOUS SYSTEM PART UNSPECIFIED 193 - MALIGNANT NEOPLASM OF THYROID GLAND 194 - MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS AND RELATED STRUCTURES 194.0 - MALIGNANT NEOPLASM OF ADRENAL GLAND 194.1 - MALIGNANT NEOPLASM OF PARATHYROID GLAND 194.3 - MALIGNANT NEOPLASM OF PITUITARY GLAND AND CRANIOPHARYNGEAL DUCT 194.4 - MALIGNANT NEOPLASM OF PINEAL GLAND 194.5 - MALIGNANT NEOPLASM OF CAROTID BODY 194.6 - MALIGNANT NEOPLASM OF AORTIC BODY AND OTHER PARAGANGLIA 194.8 - MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS AND RELATED STRUCTURES 194.9 - MALIGNANT NEOPLASM OF ENDOCRINE GLAND SITE UNSPECIFIED 195 - MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES 195.0 - MALIGNANT NEOPLASM OF HEAD FACE AND NECK 195.1 - MALIGNANT NEOPLASM OF THORAX 195.2 - MALIGNANT NEOPLASM OF ABDOMEN 195.3 - MALIGNANT NEOPLASM OF PELVIS 195.4 - MALIGNANT NEOPLASM OF UPPER LIMB 195.5 - MALIGNANT NEOPLASM OF LOWER LIMB 195.8 - MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES 196 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF LYMPH NODES 196.0 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF LYMPH NODES OF HEAD FACE AND NECK 196.1 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF INTRATHORACIC LYMPH NODES 196.2 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF INTRA-ABDOMINAL LYMPH NODES 196.3 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF LYMPH NODES OF AXILLA AND UPPER LIMB 196.5 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 196.6 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF INTRAPELVIC LYMPH NODES 196.8 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF LYMPH NODES OF MULTIPLE SITES 196.9 - SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM OF LYMPH NODES SITE UNSPECIFIED 197 - SECONDARY MALIGNANT NEOPLASM OF RESPIRATORY AND DIGESTIVE SYSTEMS 197.0 - SECONDARY MALIGNANT NEOPLASM OF LUNG 197.1 - SECONDARY MALIGNANT NEOPLASM OF MEDIASTINUM 197.2 - SECONDARY MALIGNANT NEOPLASM OF PLEURA 197.3 - SECONDARY MALIGNANT NEOPLASM OF OTHER RESPIRATORY ORGANS 197.4 - SECONDARY MALIGNANT NEOPLASM OF SMALL INTESTINE INCLUDING DUODENUM 197.5 - SECONDARY MALIGNANT NEOPLASM OF LARGE INTESTINE AND RECTUM 197.6 - SECONDARY MALIGNANT NEOPLASM OF RETROPERITONEUM AND PERITONEUM 197.7 - MALIGNANT NEOPLASM OF LIVER SECONDARY

197.8 - SECONDARY MALIGNANT NEOPLASM OF OTHER DIGESTIVE ORGANS AND SPLEEN

198 - SECONDARY MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES

198.0 - SECONDARY MALIGNANT NEOPLASM OF KIDNEY

198.1 - SECONDARY MALIGNANT NEOPLASM OF OTHER URINARY ORGANS 198.2 - SECONDARY MALIGNANT NEOPLASM OF SKIN 198.3 - SECONDARY MALIGNANT NEOPLASM OF BRAIN AND SPINAL CORD 198.4 - SECONDARY MALIGNANT NEOPLASM OF OTHER PARTS OF NERVOUS SYSTEM 198.5 - SECONDARY MALIGNANT NEOPLASM OF BONE AND BONE MARROW 198.6 - SECONDARY MALIGNANT NEOPLASM OF OVARY 198.7 - SECONDARY MALIGNANT NEOPLASM OF ADRENAL GLAND 198.8 - SECONDARY MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES 198.81 - SECONDARY MALIGNANT NEOPLASM OF BREAST 198.82 - SECONDARY MALIGNANT NEOPLASM OF GENITAL ORGANS 198.89 - SECONDARY MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES 199 - MALIGNANT NEOPLASM WITHOUT SPECIFICATION OF SITE 199.0 - DISSEMINATED MALIGNANT NEOPLASM 199.1 - OTHER MALIGNANT NEOPLASM OF UNSPECIFIED SITE 199.2 - MALIGNANT NEOPLASM ASSOCIATED WITH TRANSPLANTED ORGAN 200 - LYMPHOSARCOMA AND RETICULOSARCOMA AND OTHER SPECIFIED MALIGNANT TUMORS OF LYMPHATIC TISSUE 200.0 - RETICULOSARCOMA 200.00 - RETICULOSARCOMA UNSPECIFIED SITE 200.01 - RETICULOSARCOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 200.02 - RETICULOSARCOMA INVOLVING INTRATHORACIC LYMPH NODES 200.03 - RETICULOSARCOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 200.04 - RETICULOSARCOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 200.05 - RETICULOSARCOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 200.06 - RETICULOSARCOMA INVOLVING INTRAPELVIC LYMPH NODES 200.07 - RETICULOSARCOMA INVOLVING SPLEEN 200.08 - RETICULOSARCOMA INVOLVING LYMPH NODES OF MULTIPLE SITES 200.1 - LYMPHOSARCOMA 200.10 - LYMPHOSARCOMA UNSPECIFIED SITE 200.11 - LYMPHOSARCOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 200.12 - LYMPHOSARCOMA INVOLVING INTRATHORACIC LYMPH NODES 200.13 - LYMPHOSARCOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 200.14 - LYMPHOSARCOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 200.15 - LYMPHOSARCOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 200.16 - LYMPHOSARCOMA INVOLVING INTRAPELVIC LYMPH NODES 200.17 - LYMPHOSARCOMA INVOLVING SPLEEN 200.18 - LYMPHOSARCOMA INVOLVING LYMPH NODES OF MULTIPLE SITES 200.2 - BURKITT'S TUMOR OR LYMPHOMA 200.20 - BURKITT'S TUMOR OR LYMPHOMA UNSPECIFIED SITE 200.21 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 200.22 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING INTRATHORACIC LYMPH NODES 200.23 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 200.24 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 200.25 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 200.26 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES 200.27 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING SPLEEN 200.28 - BURKITT'S TUMOR OR LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES

| 200.3 - MARGINAL ZONE LYMPHOMA |
|---|
| 200.30 - MARGINAL ZONE LYMPHOMA UNSPECIFIED SITE |
| 200.31 - MARGINAL ZONE LYMPHOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| 200.32 - MARGINAL ZONE LYMPHOMA INVOLVING INTRATHORACIC LYMPH NODES |
| 200.33 - MARGINAL ZONE LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| 200.34 - MARGINAL ZONE LYMPHOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| 200.35 - MARGINAL ZONE LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| 200.36 - MARGINAL ZONE LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES |
| 200.37 - MARGINAL ZONE LYMPHOMA INVOLVING SPLEEN |
| 200.38 - MARGINAL ZONE LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| 200.4 - MANTLE CELL LYMPHOMA |
| 200.40 - MANTLE CELL LYMPHOMA UNSPECIFIED SITE |
| 200.41 - MANTLE CELL LYMPHOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| 200.42 - MANTLE CELL LYMPHOMA INVOLVING INTRATHORACIC LYMPH NODES |
| 200.43 - MANTLE CELL LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| 200.44 - MANTLE CELL LYMPHOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| 200.45 - MANTLE CELL LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| 200.46 - MANTLE CELL LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES |
| 200.47 - MANTLE CELL LYMPHOMA INVOLVING SPLEEN |
| 200.48 - MANTLE CELL LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| 200.5 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA |
| 200.50 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA UNSPECIFIED SITE |
| 200.51 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| 200.52 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING INTRATHORACIC LYMPH NODES |
| 200.53 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| 200.54 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| 200.55 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| 200.56 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES |
| 200.57 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING SPLEEN |
| 200.58 - PRIMARY CENTRAL NERVOUS SYSTEM LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| 200.6 - ANAPLASTIC LARGE CELL LYMPHOMA |
| 200.60 - ANAPLASTIC LARGE CELL LYMPHOMA UNSPECIFIED SITE |
| 200.61 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| 200.62 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING INTRATHORACIC LYMPH NODES |
| 200.63 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| 200.64 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| 200.65 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| 200.66 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES |
| 200.67 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING SPLEEN |
| 200.68 - ANAPLASTIC LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| 200.7 - LARGE CELL LYMPHOMA |
| 200.70 - LARGE CELL LYMPHOMA UNSPECIFIED SITE |
| 200.71 - LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| 200.72 - LARGE CELL LYMPHOMA INVOLVING INTRATHORACIC LYMPH NODES |
| 200.73 - LARGE CELL LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| 200.74 - LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |

200.75 - LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 200.76 - LARGE CELL LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES 200.77 - LARGE CELL LYMPHOMA INVOLVING SPLEEN 200.78 - LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES 200.8 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA 200.80 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA UNSPECIFIED SITE 200.81 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 200.82 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRATHORACIC LYMPH NODES 200.83 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 200.84 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 200.85 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 200.86 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRAPELVIC LYMPH NODES 200.87 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING SPLEEN 200.88 - OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF MULTIPLE SITES 201 - HODGKIN'S DISEASE 201.0 - HODGKIN'S PARAGRANULOMA 201.00 - HODGKIN'S PARAGRANULOMA UNSPECIFIED SITE 201.01 - HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.02 - HODGKIN'S PARAGRANULOMA INVOLVING INTRATHORACIC LYMPH NODES 201.03 - HODGKIN'S PARAGRANULOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.04 - HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.05 - HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.06 - HODGKIN'S PARAGRANULOMA INVOLVING INTRAPELVIC LYMPH NODES 201.07 - HODGKIN'S PARAGRANULOMA INVOLVING SPLEEN 201.08 - HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF MULTIPLE SITES 201.1 - HODGKIN'S GRANULOMA 201.10 - HODGKIN'S GRANULOMA UNSPECIFIED SITE 201.11 - HODGKIN'S GRANULOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.12 - HODGKIN'S GRANULOMA INVOLVING INTRATHORACIC LYMPH NODES 201.13 - HODGKIN'S GRANULOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.14 - HODGKIN'S GRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.15 - HODGKIN'S GRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.16 - HODGKIN'S GRANULOMA INVOLVING INTRAPELVIC LYMPH NODES 201.17 - HODGKIN'S GRANULOMA INVOLVING SPLEEN 201.18 - HODGKIN'S GRANULOMA INVOLVING LYMPH NODES OF MULTIPLE SITES 201.2 - HODGKIN'S SARCOMA 201.20 - HODGKIN'S SARCOMA UNSPECIFIED SITE 201.21 - HODGKIN'S SARCOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.22 - HODGKIN'S SARCOMA INVOLVING INTRATHORACIC LYMPH NODES 201.23 - HODGKIN'S SARCOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.24 - HODGKIN'S SARCOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.25 - HODGKIN'S SARCOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.26 - HODGKIN'S SARCOMA INVOLVING INTRAPELVIC LYMPH NODES 201.27 - HODGKIN'S SARCOMA INVOLVING SPLEEN 201.28 - HODGKIN'S SARCOMA INVOLVING LYMPH NODES OF MULTIPLE SITES

201.4 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE

201.40 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE UNSPECIFIED SITE 201.41 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.42 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING INTRATHORACIC LYMPH NODES 201.43 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.44 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.45 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.46 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING INTRAPELVIC LYMPH NODES 201.47 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING SPLEEN 201.48 - HODGKIN'S DISEASE LYMPHOCYTIC-HISTIOCYTIC PREDOMINANCE INVOLVING LYMPH NODES OF MULTIPLE SITES 201.5 - HODGKIN'S DISEASE NODULAR SCLEROSIS 201.50 - HODGKIN'S DISEASE NODULAR SCLEROSIS UNSPECIFIED SITE 201.51 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.52 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING INTRATHORACIC LYMPH NODES 201.53 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.54 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.55 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.56 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING INTRAPELVIC LYMPH NODES 201.57 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING SPLEEN 201.58 - HODGKIN'S DISEASE NODULAR SCLEROSIS INVOLVING LYMPH NODES OF MULTIPLE SITES 201.6 - HODGKIN'S DISEASE MIXED CELLULARITY 201.60 - HODGKIN'S DISEASE MIXED CELLULARITY UNSPECIFIED SITE 201.61 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.62 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING INTRATHORACIC LYMPH NODES 201.63 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.64 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.65 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.66 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING INTRAPELVIC LYMPH NODES 201.67 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING SPLEEN 201.68 - HODGKIN'S DISEASE MIXED CELLULARITY INVOLVING LYMPH NODES OF MULTIPLE SITES 201.7 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION 201.70 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION UNSPECIFIED SITE 201.71 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING LYMPH NODES OF HEAD FACE AND NECK 201.72 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING INTRATHORACIC LYMPH NODES 201.73 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING INTRA-ABDOMINAL LYMPH NODES 201.74 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB 201.75 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB 201.76 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING INTRAPELVIC LYMPH NODES 201.77 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING SPLEEN 201.78 - HODGKIN'S DISEASE LYMPHOCYTIC DEPLETION INVOLVING LYMPH NODES OF MULTIPLE SITES 201.9 - HODGKIN'S DISEASE UNSPECIFIED TYPE 201.90 - HODGKIN'S DISEASE UNSPECIFIED TYPE UNSPECIFIED SITE 201.91 - HODGKIN'S DISEASE, UNSPECIFIED TYPE, LYMPH NODES OF HEAD, FACE, AND NECK



| | | | Unmat | tched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optur | n | | Market | | | POOL | .ED | |
| Variable | Budesonide alone | Budesonide- | St. Diff. | Budesonide alone | Budesonide- | St. Diff. | Budesonide alone | Budesonide- | St. Diff. |
| | | formoterol | Jt. Dill. | | formoterol | Jt. Dill. | | formoterol | St. Dill. |
| Number of patients | 6,337 | 24,000 | | 7,38 | 0 28,864 | | 13,717 | 52,864 | |
| Year of Cohort Entry Date | | | | | | | | | |
| 2007; n (%) | 1,064 (16.8%) | 255 (1.1%) | 0.053 | 690 (9.3%) | 366 (1.3%) | 0.035 | 1,754 (12.8%) | 621 (1.2%) | 0.467 |
| 2008; n (%) | 841 (13.3%) | 968 (4.0%) | 0.032 | 559 (7.6%) | 1,296 (4.5%) | 0.013 | 1,400 (10.2%) | 2,264 (4.3%) | 0.229 |
| 2009; n (%) | 699 (11.0%) | 1,427 (5.9%) | 0.018 | 663 (9.0%) | 2,025 (7.0%) | 0.007 | 1,362 (9.9%) | 3,452 (6.5%) | 0.124 |
| 2010; n (%) | 651 (10.3%) | 1,868 (7.8%) | 0.008 | 686 (9.3%) | 2,777 (9.6%) | -0.001 | 1,337 (9.7%) | 4,645 (8.8%) | 0.031 |
| 2011; n (%) | 568 (9.0%) | 1,747 (7.3%) | 0.006 | 688 (9.3%) | 2,691 (9.3%) | 0.000 | 1,256 (9.2%) | 4,438 (8.4%) | 0.028 |
| 2012; n (%) | 497 (7.8%) | 1,832 (7.6%) | 0.001 | 763 (10.3%) | 3,144 (10.9%) | -0.002 | 1,260 (9.2%) | 4,976 (9.4%) | -0.007 |
| 2013; n (%) | 497 (7.8%) | 2,017 (8.4%) | -0.002 | 723 (9.8%) | 3,125 (10.8%) | -0.003 | 1,220 (8.9%) | 5,142 (9.7%) | -0.028 |
| 2014; n (%) | 439 (6.9%) | 1,485 (6.2%) | 0.003 | 784 (10.6%) | 4,332 (15.0%) | -0.012 | 1,223 (8.9%) | 5,817 (11.0%) | -0.070 |
| 2015; n (%) | 393 (6.2%) | 1,076 (4.5%) | 0.007 | 642 (8.7%) | 2,723 (9.4%) | -0.002 | 1,035 (7.5%) | 3,799 (7.2%) | 0.011 |
| 2016; n (%) | 250 (3.9%) | 2,197 (9.2%) | -0.021 | 493 (6.7%) | 2,082 (7.2%) | -0.002 | 743 (5.4%) | 4,279 (8.1%) | -0.108 |
| 2017; n (%) | 143 (2.3%) | 2,112 (8.8%) | -0.028 | 379 (5.1%) | 1,780 (6.2%) | -0.005 | 522 (3.8%) | 3,892 (7.4%) | -0.157 |
| 2018; n (%) | 130 (2.1%) | 2,606 (10.9%) | -0.035 | 310 (4.2%) | 2,523 (8.7%) | -0.018 | 440 (3.2%) | 5,129 (9.7%) | -0.267 |
| 2019; n (%) | 121 (1.9%) | 2,779 (11.6%) | -0.037 | NA | NA | NA | NA | NA | NA |
| 2020; n (%) | 44 (0.7%) | 1,631 (6.8%) | -0.032 | NA | NA | NA | NA | NA | NA |
| Age | | | | | | | | | |
| mean (sd) | 42.71 (20.00) | 51.86 (19.19) | -0.467 | 43.92 (20.01) | 48.36 (17.11) | -0.238 | 43.36 (20.01) | 49.95 (18.08) | -0.346 |
| median [IQR] | 43.00 [27.00, 58.00] | 54.00 [39.00, 67.00] | -0.561 | 47.00 [27.00, 59.00] | 51.00 [39.00, 60.00] | -0.215 | 45.15 (20.01) | 52.36 (18.08) | -0.378 |
| Age categories | | (, | | . , . | . , . | | , , | , , | |
| 12-17; n (%) | 1,167 (18.4%) | 1,752 (7.3%) | 0.031 | 1,275 (17.3%) | 2,255 (7.8%) | 0.027 | 2,442 (17.8%) | 4,007 (7.6%) | 0.310 |
| 18-39; n (%) | 1,616 (25.5%) | 4,397 (18.3%) | 0.015 | 1,641 (22.2%) | 5,370 (18.6%) | 0.008 | 3,257 (23.7%) | 9,767 (18.5%) | 0.128 |
| 40 - 64; n (%) | 2,590 (40.9%) | 10,603 (44.2%) | -0.005 | 3,478 (47.1%) | 17,391 (60.3%) | -0.018 | 6,068 (44.2%) | 27,994 (53.0%) | -0.177 |
| >= 65; n (%) | 964 (15.2%) | 7,248 (30.2%) | -0.032 | 986 (13.4%) | 3,848 (13.3%) | 0.000 | 1,950 (14.2%) | 11,096 (21.0%) | -0.179 |
| Geographic Region | 33 . (23.270) | 7,210 (50.270) | 0.002 | 500 (25.170) | 0,010 (10.070) | 0.000 | 1,550 (1/5) | 11,030 (21.070) | 0.275 |
| Northeast; n (%) | 916 (14.5%) | 2,632 (11.0%) | 0.010 | 1,649 (22.3%) | 5,792 (20.1%) | 0.005 | 2,565 (18.7%) | 8,424 (15.9%) | 0.074 |
| South; n (%) | 2,191 (34.6%) | 10,968 (45.7%) | -0.018 | 2,151 (29.1%) | 11,533 (40.0%) | -0.019 | 4,342 (31.7%) | 22,501 (42.6%) | -0.227 |
| Midwest; n (%) | 1,960 (30.9%) | 5,075 (21.1%) | 0.019 | 2,404 (32.6%) | 7,125 (24.7%) | 0.015 | 4,364 (31.8%) | 12,200 (23.1%) | 0.196 |
| West; n (%) | 1,270 (20.0%) | 5,325 (22.2%) | -0.005 | 1,118 (15.1%) | 4,153 (14.4%) | 0.002 | 2,388 (17.4%) | 9,478 (17.9%) | -0.013 |
| Unknown/Missing; n (%) | 1,270 (20.0%)<br>NA | NA | NA | 58 (0.8%) | 261 (0.9%) | -0.001 | 2,366 (17.470)<br>NA | NA | NA |
| Metropolitan Statistical Area | NA . | INA | INA | 36 (0.6%) | 201 (0.9%) | -0.001 | INA | NA | IVA |
| <u> </u> | NA | NA | NIA | C 0C0 (02 20/) | 22 002 /70 00/\ | 0.004 | NA | NA | NA |
| Urban; n (%) | | | NA | 6,069 (82.2%) | 22,803 (79.0%) | | | | |
| Rural; n (%) | NA<br>NA | NA | NA | 108 (1.5%) | 705 (2.4%) | -0.006 | NA | NA | NA |
| Unknown/Missing; n (%) | NA | NA | NA | 1,203 (16.3%) | 5,356 (18.6%) | -0.006 | NA | NA | NA |
| General Health Related Measures | 12 (0.2%) | 24.5 (0.00() | 0.000 | 20 (0.40() | 427 (0.40() | 0.000 | 0.42 (0.20() | 2.42 (0.6%) | 0.045 |
| Alcohol/Drug abuse or dependence; n (%) | 12 (0.2%) | 216 (0.9%) | -0.009 | 30 (0.4%) | 127 (0.4%) | 0.000 | 042 (0.3%) | 343 (0.6%) | -0.045 |
| Obesity or Overweight; n (%) | 333 (5.3%) | 3,464 (14.4%) | -0.029 | 440 (6.0%) | 2,772 (9.6%) | -0.013 | 773 (5.6%) | 6,236 (11.8%) | -0.221 |
| Obesity; n (%) | 269 (4.2%) | 2,786 (11.6%) | -0.026 | 376 (5.1%) | 2,344 (8.1%) | -0.012 | 645 (4.7%) | 5,130 (9.7%) | -0.194 |
| Overweight; n (%) | 66 (1.0%) | 798 (3.3%) | -0.016 | 74 (1.0%) | 511 (1.8%) | -0.007 | 140 (1.0%) | 1,309 (2.5%) | -0.115 |
| Cardiovascular Measures | | | | | | | | | |
| Hypertension; n (%) | 1,467 (23.1%) | 9,667 (40.3%) | -0.031 | 1,708 (23.1%) | 9,051 (31.4%) | -0.016 | 3,175 (23.1%) | 18,718 (35.4%) | -0.273 |
| Hyperlipidemia; n (%) | 1,280 (20.2%) | 7,113 (29.6%) | -0.019 | 1,309 (17.7%) | 6,483 (22.5%) | -0.011 | 2,589 (18.9%) | 13,596 (25.7%) | -0.164 |
| MI, angina, Coronary atherosclerosis and other forms of chronic | 199 (3.1%) | 1,404 (5.9%) | -0.013 | 243 (3.3%) | 1,231 (4.3%) | -0.005 | 442 (3.2%) | 2,635 (5.0%) | -0.091 |
| ischemic heart disease; n (%) | | | | • | | | | | |
| Old MI; n (%) | 22 (0.3%) | 140 (0.6%) | -0.004 | 20 (0.3%) | 78 (0.3%) | 0.000 | 042 (0.3%) | 218 (0.4%) | -0.017 |
| Acute MI; n (%) | 8 (0.1%) | 51 (0.2%) | -0.003 | 11 (0.1%) | 48 (0.2%) | -0.003 | 019 (0.1%) | 099 (0.2%) | -0.026 |
| Stable angina; n (%) | 27 (0.4%) | 277 (1.2%) | -0.009 | 29 (0.4%) | 207 (0.7%) | -0.004 | 056 (0.4%) | 484 (0.9%) | -0.062 |
| Coronary atherosclerosis and other forms of chronic ischemic | | | -0.012 | 204 (2.8%) | 1,045 (3.6%) | -0.004 | 383 (2.8%) | 2,264 (4.3%) | -0.081 |
| heart disease; n (%) | 179 (2.8%) | 1,219 (5.1%) | | | | | | | |
| History of CABG or PTCA; n (%) | 32 (0.5%) | 250 (1.0%) | -0.006 | 20 (0.3%) | 124 (0.4%) | -0.002 | 052 (0.4%) | 374 (0.7%) | -0.041 |

| Construction disease (Chapter TIA Late officially at (01) | 20 (0.50() | 224 (4.22() | 0.007 | (2 (0 00() | 270 (0.00() | 0.004 | 400 (0.70/) | E04 (4 40/) | 0.043 |
|---|---|---|---|---|---|---|---|---|---|
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%)<br>Stroke (Ischemic or hemorrhagic); n (%) | 38 (0.6%)<br>19 (0.3%) | 321 (1.3%)<br>157 (0.7%) | -0.007<br>-0.006 | 62 (0.8%)<br>26 (0.4%) | 270 (0.9%)<br>148 (0.5%) | -0.001<br>-0.001 | 100 (0.7%)<br>045 (0.3%) | 591 (1.1%)<br>305 (0.6%) | -0.042<br>-0.045 |
| TIA; n (%) | 14 (0.2%) | 127 (0.5%) | -0.005 | 33 (0.4%) | 113 (0.4%) | 0.000 | 047 (0.3%) | 240 (0.5%) | -0.032 |
| Late effects of cerebrovascular disease; n (%) | 10 (0.2%) | 102 (0.4%) | -0.004 | 12 (0.2%) | 62 (0.2%) | 0.000 | 022 (0.2%) | 164 (0.3%) | -0.020 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%) | 229 (3.6%) | 1,188 (5.0%) | -0.007 | 337 (4.6%) | 1,045 (3.6%) | 0.005 | 566 (4.1%) | 2,233 (4.2%) | -0.005 |
| Atrial fibrillation; n (%) | 108 (1.7%) | 639 (2.7%) | -0.007 | 169 (2.3%) | 460 (1.6%) | 0.005 | 277 (2.0%) | 1,099 (2.1%) | -0.007 |
| Other cardiac dysrhythmia; n (%) | 155 (2.4%) | 978 (4.1%) | -0.009 | 223 (3.0%) | 776 (2.7%) | 0.003 | 378 (2.8%) | 1,754 (3.3%) | -0.029 |
| Diabetes Related Measures | 133 (2.470) | 378 (4.176) | 0.003 | 223 (3.070) | 770 (2.770) | 0.002 | 370 (2.0%) | 1,754 (5.570) | 0.023 |
| Diabetes with or w/o complications; n (%) | 447 (7.1%) | 3,349 (14.0%) | -0.021 | 520 (7.0%) | 3,147 (10.9%) | -0.013 | 967 (7.0%) | 6,496 (12.3%) | -0.180 |
| Diabetes mellitus without mention of complications; n (%) | 430 (6.8%) | 3,099 (12.9%) | -0.019 | 485 (6.6%) | 2,986 (10.3%) | -0.013 | 915 (6.7%) | 6,085 (11.5%) | -0.167 |
| Diabetes with specified complications; n (%) | 75 (1.2%) | 814 (3.4%) | -0.015 | 87 (1.2%) | 489 (1.7%) | -0.004 | 162 (1.2%) | 1,303 (2.5%) | -0.097 |
| Diabetes with unspecified complications; n (%) | 17 (0.3%) | 151 (0.6%) | -0.004 | 17 (0.2%) | 126 (0.4%) | -0.004 | 034 (0.2%) | 277 (0.5%) | -0.051 |
| GI Conditions | 17 (0.570) | 131 (0.070) | | () | (0) | | (0.2,2,7 | | |
| GERD; n (%) | 559 (8.8%) | 3,512 (14.6%) | -0.017 | 606 (8.2%) | 3,258 (11.3%) | -0.010 | 1,165 (8.5%) | 6,770 (12.8%) | -0.140 |
| Upper GI (Diseases of esophagus, stomach and duodenum including | 333 (8.670) | 3,312 (1 110/0) | | | | | | | |
| GERD); n (%) | 698 (11.0%) | 4,098 (17.1%) | -0.016 | 788 (10.7%) | 4,062 (14.1%) | -0.010 | 1,486 (10.8%) | 8,160 (15.4%) | -0.137 |
| GI bleeding; n (%) | 78 (1.2%) | 339 (1.4%) | -0.002 | 84 (1.1%) | 392 (1.4%) | -0.003 | 162 (1.2%) | 731 (1.4%) | -0.018 |
| Non-infective enteritis and colitis; n (%) | 189 (3.0%) | 757 (3.2%) | -0.001 | 238 (3.2%) | 952 (3.3%) | -0.001 | 427 (3.1%) | 1,709 (3.2%) | -0.006 |
| Intraoperative and postprocedural complications and disorders of | | | 0.003 | 00 (4.49/) | 264 (4.20() | 0.002 | 166 (1 20/) | CEO (4. 20/) | 0.000 |
| digestive system; n (%) | 86 (1.4%) | 297 (1.2%) | 0.002 | 80 (1.1%) | 361 (1.3%) | -0.002 | 166 (1.2%) | 658 (1.2%) | 0.000 |
| Disorders of gallbladder, biliary tract and pancreas; n (%) | 50 (0.8%) | 264 (1.1%) | -0.003 | 61 (0.8%) | 283 (1.0%) | -0.002 | 111 (0.8%) | 547 (1.0%) | -0.021 |
| Rheumatic Conditions | | | | | | | | | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n | 68 (1.1%) | 405 (1.7%) | -0.005 | 108 (1.5%) | 414 (1.4%) | 0.001 | 176 (1.3%) | 819 (1.5%) | -0.017 |
| (%) | | | | | | | | | |
| Osteoarthrosis; n (%) | 405 (6.4%) | 2,814 (11.7%) | -0.018 | 562 (7.6%) | 2,559 (8.9%) | -0.005 | 967 (7.0%) | 5,373 (10.2%) | -0.114 |
| Other rheumatic disorders (including gout); n (%) | 1,177 (18.6%) | 6,074 (25.3%) | -0.014 | 1,481 (20.1%) | 6,665 (23.1%) | -0.006 | 2,658 (19.4%) | 12,739 (24.1%) | -0.114 |
| Gout and other crystal arthropathies; n (%) | 37 (0.6%) | 359 (1.5%) | -0.009 | 40 (0.5%) | 294 (1.0%) | -0.006 | 077 (0.6%) | 653 (1.2%) | -0.064 |
| Other rheumatic disorders; n (%) | 1,156 (18.2%) | 5,834 (24.3%) | -0.013 | 1,455 (19.7%) | 6,470 (22.4%) | -0.006 | 2,611 (19.0%) | 12,304 (23.3%) | -0.105 |
| Neuro Conditions | | | | | | | | | |
| Alzheimer and other Dementia Disease; n (%) | 37 (0.6%) | 276 (1.1%) | -0.005 | 34 (0.5%) | 141 (0.5%) | 0.000 | 071 (0.5%) | 417 (0.8%) | -0.037 |
| Seizure disorders (epilepsy); n (%) | 30 (0.5%) | 158 (0.7%) | -0.003 | 40 (0.5%) | 164 (0.6%) | -0.001 | 070 (0.5%) | 322 (0.6%) | -0.014 |
| Delirium/Psychosis; n (%) | 50 (0.8%) | 228 (0.9%) | -0.001 | 46 (0.6%) | 175 (0.6%) | 0.000 | 096 (0.7%) | 403 (0.8%) | -0.012 |
| Other Conditions | (() | | | () | | | | // | |
| Hypothyroidism; n (%) | 550 (8.7%) | 2,811 (11.7%) | -0.009 | 552 (7.5%) | 2,594 (9.0%) | -0.005 | 1,102 (8.0%) | 5,405 (10.2%) | -0.077 |
| Chronic kidney disease stages I-III; n (%) | 100 (1.6%) | 1,021 (4.3%) | -0.016 | 61 (0.8%) | 422 (1.5%) | -0.007 | 161 (1.2%) | 1,443 (2.7%) | -0.109 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 31 (0.5%) | 229 (1.0%) | -0.006 | 20 (0.3%) | 121 (0.4%) | -0.002 | 051 (0.4%) | 350 (0.7%) | -0.041 |
| COPD; n (%) | 283 (4.5%) | 2,954 (12.3%) | -0.027 | 381 (5.2%) | 2,608 (9.0%) | -0.014 | 664 (4.8%) | 5,562 (10.5%) | -0.216 |
| Obstructive sleep apnea; n (%) | 302 (4.8%) | 2,390 (10.0%) | -0.019<br>-0.002 | 378 (5.1%) | 2,438 (8.4%) | -0.013<br>-0.001 | 680 (5.0%) | 4,828 (9.1%) | -0.161<br>-0.019 |
| Syncope; n (%) Falls; n (%) | 67 (1.1%)<br>67 (1.1%) | 319 (1.3%)<br>422 (1.8%) | -0.002<br>-0.006 | 75 (1.0%)<br>39 (0.5%) | 315 (1.1%)<br>174 (0.6%) | -0.001 | 142 (1.0%)<br>106 (0.8%) | 634 (1.2%)<br>596 (1.1%) | -0.019 |
| VTE; n (%) | 35 (0.6%) | 200 (0.8%) | -0.006 | 61 (0.8%) | 266 (0.9%) | -0.001 | 096 (0.7%) | 466 (0.9%) | -0.031 |
| Combined comorbidity score, 365 days | 33 (0.6%) | 200 (0.8%) | -0.002 | 61 (0.6%) | 200 (0.9%) | -0.001 | 096 (0.7%) | 466 (0.9%) | -0.022 |
| | 1.14 (0.91) | 1.38 (1.37) | -0.206 | 1 15 (0 90) | 1.14 (0.97) | 0.011 | 1 15 (0 00) | 1 25 /1 17\ | -0.096 |
| mean (sd)median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 2.00] | 0.000 | 1.15 (0.89)<br>1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.000 | 1.15 (0.90)<br>1.00 (0.90) | 1.25 (1.17)<br>1.00 (1.17) | 0.000 |
| Frailty Score: Empirical Version 365 days as Categories | 1.00 [1.00, 1.00] | 1.00 [1.00, 2.00] | 0.000 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.000 | 1.00 (0.50) | 1.00 (1.17) | 0.000 |
| <0.1 non frail; n (%) | 4,334 (68.4%) | 16,797 (70.0%) | -0.002 | 4,405 (59.7%) | 15,841 (54.9%) | 0.006 | 8,739 (63.7%) | 32,638 (61.7%) | 0.041 |
| 0.1 -<0.2 prefrail; n (%) | 1,342 (21.2%) | 4,099 (17.1%) | 0.002 | 1,854 (25.1%) | 7,413 (25.7%) | -0.001 | 3,196 (23.3%) | 11,512 (21.8%) | 0.036 |
| > 0.2 frail; n (%) | 661 (10.4%) | 3,104 (12.9%) | -0.007 | 1,121 (15.2%) | 5,610 (19.4%) | -0.010 | 1,782 (13.0%) | 8,714 (16.5%) | -0.099 |
| Medication Use | 001 (10.470) | 3,104 (12.370) | 0.007 | 1,121 (13.270) | 3,010 (13.470) | 0.010 | 1,702 (13.070) | 0,714 (10.570) | 0.033 |
| Use of oral corticosteroids; n (%) | 2,830 (44.7%) | 13,878 (57.8%) | -0.018 | 7,014 (95.0%) | 27,411 (95.0%) | 0.000 | 9,844 (71.8%) | 41,289 (78.1%) | -0.146 |
| Use of antidepressants; n (%) | 1,161 (18.3%) | 6,021 (25.1%) | -0.015 | 1,607 (21.8%) | 7,480 (25.9%) | -0.008 | 2,768 (20.2%) | 13,501 (25.5%) | -0.126 |
| Use of anticonvulsants; n (%) | 339 (5.3%) | 2,529 (10.5%) | -0.013 | 536 (7.3%) | 2,666 (9.2%) | -0.008 | 875 (6.4%) | 5,195 (9.8%) | -0.125 |
| 050 0. 00011441541165, 11 (70) | | | | | | | | 7,124 (13.5%) | -0.123 |
| Use of beta blocker OR calcium channel blocker: n (%) | 579 (9 1%) | 3.575 (14 9%) | -0.017 | 803 (10 4%) | | | | | |
| Use of beta blocker OR calcium channel blocker; n (%)<br>Use of PPIs; n (%) | 579 (9.1%)<br>870 (13.7%) | 3,575 (14.9%)<br>5,203 (21.7%) | -0.017<br>-0.019 | 803 (10.9%)<br>1,526 (20.7%) | 3,549 (12.3%)<br>7,048 (24.4%) | -0.004<br>-0.008 | 1,382 (10.1%)<br>2,396 (17.5%) | 12,251 (23.2%) | -0.142 |

| | - | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Use of antipsychotics; n (%) | 83 (1.3%) | 527 (2.2%) | -0.007 | 107 (1.4%) | 534 (1.9%) | -0.004 | 190 (1.4%) | 1,061 (2.0%) | -0.046 |
| Use of anxiolytics/hypnotics; n (%) | 329 (5.2%) | 1,814 (7.6%) | -0.009 | 486 (6.6%) | 2,517 (8.7%) | -0.008 | 815 (5.9%) | 4,331 (8.2%) | -0.090 |
| Use of dementia meds; n (%) | 23 (0.4%) | 220 (0.9%) | -0.006 | 26 (0.4%) | 122 (0.4%) | 0.000 | 049 (0.4%) | 342 (0.6%) | -0.028 |
| Use of antiparkinsonian meds; n (%) | 58 (0.9%) | 448 (1.9%) | -0.008 | 104 (1.4%) | 519 (1.8%) | -0.003 | 162 (1.2%) | 967 (1.8%) | -0.049 |
| Use of Benzodiazepine; n (%) | 541 (8.5%) | 2,733 (11.4%) | -0.009 | 880 (11.9%) | 3,889 (13.5%) | -0.004 | 1,421 (10.4%) | 6,622 (12.5%) | -0.066 |
| All antidiabetic medications; n (%) | 351 (5.5%) | 2,778 (11.6%) | -0.021 | 499 (6.8%) | 2,817 (9.8%) | -0.010 | 850 (6.2%) | 5,595 (10.6%) | -0.159 |
| ACEI/ARB; n (%) | 996 (15.7%) | 6,682 (27.8%) | -0.026 | 1,410 (19.1%) | 7,124 (24.7%) | -0.012 | 2,406 (17.5%) | 13,806 (26.1%) | -0.209 |
| Use of Anticoagulants; n (%) | 116 (1.8%) | 674 (2.8%) | -0.007 | 165 (2.2%) | 608 (2.1%) | 0.001 | 281 (2.0%) | 1,282 (2.4%) | -0.027 |
| Use of Amiodarone; n (%) | 11 (0.2%) | 55 (0.2%) | 0.000 | 17 (0.2%) | 44 (0.2%) | 0.000 | 028 (0.2%) | 099 (0.2%) | 0.000 |
| Digoxin; n (%) | 26 (0.4%) | 100 (0.4%) | 0.000 | 45 (0.6%) | 114 (0.4%) | 0.003 | 071 (0.5%) | 214 (0.4%) | 0.015 |
| Use of Diuretics; n (%) | 813 (12.8%) | 5,229 (21.8%) | -0.022 | 1,183 (16.0%) | 5,938 (20.6%) | -0.011 | 1,996 (14.6%) | 11,167 (21.1%) | -0.170 |
| Use of Aspirin; n (%) | 21 (0.3%) | 110 (0.5%) | -0.003 | 26 (0.4%) | 144 (0.5%) | -0.001 | 047 (0.3%) | 254 (0.5%) | -0.032 |
| NSAIDs (NOT including aspirin); n (%) | 533 (8.4%) | 3,311 (13.8%) | -0.016 | 861 (11.7%) | 4,372 (15.1%) | -0.009 | 1,394 (10.2%) | 7,683 (14.5%) | -0.131 |
| HRT (Use of estrogens, progestins, androgens); n (%) | 889 (14.0%) | 2,782 (11.6%) | 0.007 | 1,178 (16.0%) | 4,006 (13.9%) | 0.005 | 2,067 (15.1%) | 6,788 (12.8%) | 0.066 |
| Use of Statins ; n (%) | 1,037 (16.4%) | 6,365 (26.5%) | -0.022 | 1,290 (17.5%) | 6,323 (21.9%) | -0.010 | 2,327 (17.0%) | 12,688 (24.0%) | -0.174 |
| Healthcare Utilization Measures | | | | | | | | | |
| Use of any drugs claims | | | | | | | | | |
| mean (sd) | 22.04 (17.13) | 26.38 (19.37) | -0.237 | 24.69 (17.07) | 27.04 (18.47) | -0.132 | 23.47 (17.10) | 26.74 (18.88) | -0.182 |
| median [IQR] | 18.00 [10.00, 29.00] | 22.00 [12.00, 35.00] | -0.219 | 21.00 [12.00, 33.00] | 23.00 [14.00, 36.00] | -0.112 | 19.61 (17.10) | 22.55 (18.88) | -0.163 |
| Number of office visits | | | | | | | | | |
| mean (sd) | 9.78 (7.99) | 11.67 (9.61) | -0.214 | 11.12 (8.19) | 11.44 (7.91) | -0.040 | 10.50 (8.10) | 11.54 (8.72) | -0.124 |
| median [IQR] | 8.00 [5.00, 12.00] | 9.00 [5.00, 15.00] | -0.113 | 9.00 [6.00, 14.00] | 10.00 [6.00, 15.00] | -0.124 | 8.54 (8.10) | 9.55 (8.72) | -0.120 |
| Number of ED visits | | | | | | | | | |
| mean (sd) | 0.31 (0.75) | 0.45 (1.08) | -0.151 | 0.52 (1.14) | 0.56 (1.20) | -0.034 | 0.42 (0.98) | 0.51 (1.15) | -0.084 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (0.98) | 0.00 (1.15) | 0.000 |
| Number of hospitalizations | | | | | | | | | |
| mean (sd) | 0.02 (0.19) | 0.04 (0.27) | -0.086 | 0.16 (1.28) | 0.17 (1.23) | -0.008 | 0.10 (0.95) | 0.11 (0.93) | -0.011 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (0.95) | 0.00 (0.93) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 14 (0.2%) | 152 (0.6%) | -0.006 | 40 (0.5%) | 186 (0.6%) | -0.001 | 054 (0.4%) | 338 (0.6%) | -0.028 |
| Old hospitalizations (-365 to -31 days); n (%) | 354 (5.6%) | 1,508 (6.3%) | -0.003 | 503 (6.8%) | 1,972 (6.8%) | 0.000 | 857 (6.2%) | 3,480 (6.6%) | -0.016 |
| Number of Pulmonologist/Allergist visits | | | | | | | | | |
| mean (sd) | 0.02 (0.23) | 0.04 (0.43) | -0.058 | 1.37 (3.61) | 1.35 (3.58) | 0.006 | 0.75 (2.65) | 0.76 (2.66) | -0.004 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (2.65) | 0.00 (2.66) | 0.000 |
| Pulmonologist /allergist on CED; n (%) | 3 (0.0%) | 61 (0.3%) | -0.008 | 465 (6.3%) | 2,178 (7.5%) | -0.005 | 468 (3.4%) | 2,239 (4.2%) | -0.042 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 0.18 (2.69) | 0.28 (2.91) | -0.036 | 0.16 (1.28) | 0.17 (1.23) | -0.008 | 0.17 (2.06) | 0.22 (2.16) | -0.024 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (2.06) | 0.00 (2.16) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood chemistry | 1,597 (25.2%) | 9,025 (37.6%) | -0.022 | 1,762 (23.9%) | 8,401 (29.1%) | -0.010 | 3,359 (24.5%) | 17,426 (33.0%) | -0.189 |
| test; n (%) | 2,557 (25.270) | 3)023 (371070) | 0.022 | 2)702 (20.370) | 0) 101 (2311/0) | 0.010 | 0,000 (2 11070) | 17,120 (33.070) | 0.105 |
| Number of HbA1C test ordered | | | | | | | | | |
| mean (sd) | 0.29 (0.82) | 0.62 (1.17) | -0.327 | 0.28 (0.77) | 0.40 (0.94) | -0.140 | 0.28 (0.79) | 0.50 (1.05) | -0.237 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (0.79) | 0.00 (1.05) | 0.000 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; | 194 (3.1%) | 890 (3.7%) | -0.003 | 250 (3.4%) | 1,119 (3.9%) | -0.003 | 444 (3.2%) | 2,009 (3.8%) | -0.033 |
| n (%) | | | | | | | | | |
| Number of Mammograms (Breast cancer screening); n (%) | 849 (13.4%) | 3,434 (14.3%) | -0.002 | 993 (13.5%) | 3,999 (13.9%) | -0.001 | 1,842 (13.4%) | 7,433 (14.1%) | -0.020 |
| Number of Pap smear (Cervical cancer screening); n (%) | 898 (14.2%) | 2,170 (9.0%) | 0.015 | 1,035 (14.0%) | 3,178 (11.0%) | 0.008 | 1,933 (14.1%) | 5,348 (10.1%) | 0.123 |
| Flu vaccine; n (%) | 1,130 (17.8%) | 4,320 (18.0%) | 0.000 | 1,247 (16.9%) | 4,546 (15.7%) | 0.003 | 2,377 (17.3%) | 8,866 (16.8%) | 0.013 |
| Pneumococcal vaccine; n (%) | 325 (5.1%) | 3,234 (13.5%) | -0.028 | 449 (6.1%) | 2,077 (7.2%) | -0.004 | 774 (5.6%) | 5,311 (10.0%) | -0.165 |
| Copay for pharmacy cost (charges in U.S. \$) | | | | | | | | | |
| mean (sd) | 35.24 (31.61) | 35.92 (35.15) | -0.020 | 25.32 (23.84) | 25.69 (25.62) | -0.015 | 29.90 (27.70) | 30.33 (30.32) | -0.015 |
| median [IQR] | 29.02 [16.72, 45.16] | 29.15 [15.10, 46.93] | -0.004 | 21.25 [9.74, 34.71] | 20.90 [10.28, 34.52] | 0.014 | 24.84 (27.70) | 24.65 (30.32) | 0.007 |
| Business Type | 5 500 (25 25) | 46.005 (22.22) | 0.0 | | | | | | |
| Commercial; n (%) | 5,566 (87.8%) | 16,395 (68.3%) | 0.022 | NA | NA | NA | NA | NA | NA |
| Medicare; n (%) | 771 (12.2%) | 7,605 (31.7%) | -0.042 | NA | NA | NA | NA | NA | NA |
| Insurance Plan Type | | | | | | | | | |

| Comprehensive; n (%) | NA | NA | NA | 601 (8.1%) | 2,299 (8.0%) | 0.000 | NA | NA | NA |
|---|---|---|---|---|---|---|---|---|---|
| HMO; n (%) | NA | NA | NA | 978 (13.3%) | 3,421 (11.9%) | 0.004 | NA | NA | NA |
| PPO; n (%) | NA | NA | NA | 4,270 (57.9%) | 16,728 (58.0%) | 0.000 | NA | NA | NA |
| Others; n (%) | NA | NA | NA | 1,531 (20.7%) | 6,416 (22.2%) | -0.003 | NA | NA | NA |
| SABA; n (%) | 3,308 (52.2%) | 12,697 (52.9%) | -0.001 | 4,699 (63.7%) | 18,511 (64.1%) | -0.001 | 8,007 (58.4%) | 31,208 (59.0%) | -0.012 |
| SAMA; n (%) | 95 (1.5%) | 450 (1.9%) | -0.003 | 204 (2.8%) | 744 (2.6%) | 0.001 | 299 (2.2%) | 1,194 (2.3%) | -0.007 |
| SABA/SAMA; n (%) | 116 (1.8%) | 835 (3.5%) | -0.010 | 269 (3.6%) | 1,517 (5.3%) | -0.008 | 385 (2.8%) | 2,352 (4.4%) | -0.086 |
| ICS without budesonide; n (%) | 1,922 (30.3%) | 6,879 (28.7%) | 0.003 | 2,746 (37.2%) | 10,504 (36.4%) | 0.001 | 4,668 (34.0%) | 17,383 (32.9%) | 0.023 |
| LABA; n (%) | 493 (7.8%) | 240 (1.0%) | 0.032 | 502 (6.8%) | 447 (1.5%) | 0.026 | 995 (7.3%) | 687 (1.3%) | 0.299 |
| LAMA; n (%) | 126 (2.0%) | 1,049 (4.4%) | -0.013 | 248 (3.4%) | 1,685 (5.8%) | -0.011 | 374 (2.7%) | 2,734 (5.2%) | -0.129 |
| ICS/LABA (without budesonide-formoterol); n (%) | 635 (10.0%) | 3,591 (15.0%) | -0.014 | 825 (11.2%) | 5,565 (19.3%) | -0.021 | 1,460 (10.6%) | 9,156 (17.3%) | -0.194 |
| Blood eosinophilia test ; n (%) | 26 (0.4%) | 53 (0.2%) | 0.004 | 14 (0.2%) | 88 (0.3%) | -0.002 | 040 (0.3%) | 141 (0.3%) | 0.000 |
| Serum immunoglobulin E (IgE) level test; n (%) | 72 (1.1%) | 346 (1.4%) | -0.003 | 121 (1.6%) | 659 (2.3%) | -0.005 | 193 (1.4%) | 1,005 (1.9%) | -0.039 |
| H2 blocker; n (%) | 59 (0.9%) | 649 (2.7%) | -0.013 | 233 (3.2%) | 982 (3.4%) | -0.001 | 292 (2.1%) | 1,631 (3.1%) | -0.063 |
| Oxygen codes; n (%) | 15 (0.2%) | 156 (0.7%) | -0.007 | 37 (0.5%) | 226 (0.8%) | -0.004 | 052 (0.4%) | 382 (0.7%) | -0.041 |
| Respiratory arrest/dependence on oxygen; n (%) | 1 (0.0%) | 6 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 001 (0.0%) | 006 (0.0%) | #DIV/0! |

 $A etion link to Optum results: https://bwh-dope.aetion.com/projects/details/1657/rwrs/68456\\ A etion link to Marketscan results: https://bwh-dope.aetion.com/projects/details/1656/rwrs/68455\\$ 

| | | PS-m | natched | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optun | 1 | | Markets | scan | | POOLED | | |
| Variable | Budesonide alone | Budesonide-<br>formoterol | St. Diff. | Budesonide alone | Budesonide-<br>formoterol | St. Diff. | Budesonide<br>alone | Budesonide-<br>formoterol | St. Diff. |
| Number of patients | 5,198 | 5,198 | ; | 6,95 | 9 6,959 | | 12,157 | 12,157 | |
| Year of Cohort Entry Date | | | | | | | | | |
| 2007; n (%) | 250 (4.8%) | 245 (4.7%) | 0.0005 | 336 (4.8%) | 330 (4.7%) | 0.0005 | 586 (4.8%) | 575 (4.7%) | 0.005 |
| 2008; n (%) | 627 (12.1%) | 656 (12.6%) | -0.0014 | 521 (7.5%) | 529 (7.6%) | -0.0004 | 1,148 (9.4%) | 1,185 (9.7%) | -0.010 |
| 2009; n (%) | 647 (12.4%) | 658 (12.7%) | -0.0008 | 648 (9.3%) | 668 (9.6%) | -0.0010 | 1,295 (10.7%) | 1,326 (10.9%) | -0.006 |
| 2010; n (%) | 636 (12.2%) | 625 (12.0%) | 0.0006 | 680 (9.8%) | 692 (9.9%) | -0.0003 | 1,316 (10.8%) | 1,317 (10.8%) | 0.000 |
| 2011; n (%) | 552 (10.6%) | 538 (10.4%) | 0.0006 | 687 (9.9%) | 711 (10.2%) | -0.0009 | 1,239 (10.2%) | 1,249 (10.3%) | -0.003 |
| 2012; n (%) | 494 (9.5%) | 518 (10.0%) | -0.0016 | 761 (10.9%) | 756 (10.9%) | 0.0000 | 1,255 (10.3%) | 1,274 (10.5%) | -0.007 |
| 2013; n (%) | 496 (9.5%) | 463 (8.9%) | 0.0020 | 723 (10.4%) | 685 (9.8%) | 0.0019 | 1,219 (10.0%) | 1,148 (9.4%) | 0.020 |
| 2014; n (%) | 435 (8.4%) | 444 (8.5%) | -0.0003 | 783 (11.3%) | 793 (11.4%) | -0.0003 | 1,218 (10.0%) | 1,237 (10.2%) | -0.007 |
| 2015; n (%) | 373 (7.2%) | 356 (6.8%) | 0.0015 | 641 (9.2%) | 644 (9.3%) | -0.0003 | 1,014 (8.3%) | 1,000 (8.2%) | 0.004 |
| 2016; n (%) | 250 (4.8%) | 242 (4.7%) | 0.0005 | 491 (7.1%) | 469 (6.7%) | 0.0015 | 741 (6.1%) | 711 (5.8%) | 0.013 |
| 2017; n (%) | 143 (2.8%) | 151 (2.9%) | -0.0006 | 378 (5.4%) | 397 (5.7%) | -0.0013 | 521 (4.3%) | 548 (4.5%) | -0.010 |
| 2018; n (%) | 130 (2.5%) | 146 (2.8%) | -0.0018 | 310 (4.5%) | 285 (4.1%) | 0.0019 | 440 (3.6%) | 431 (3.5%) | 0.005 |
| 2019; n (%) | 121 (2.3%) | 117 (2.3%) | 0.0000 | NA | NA | NA | NA | NA | NA |
| 2020; n (%) | 44 (0.8%) | 39 (0.8%) | 0.0000 | NA | NA | NA | NA | NA. | NA |
| Age* | 44 (0.870) | 33 (0.070) | 0.0000 | 14/1 | 1471 | 1471 | 1471 | 10.1 | 1471 |
| mean (sd) | 43.68 (20.21) | 43.29 (19.29) | 0.0197 | 43.76 (19.95) | 43.63 (18.37) | 0.0068 | 43.73 (20.06) | 43.48 (18.77) | 0.013 |
| median [IQR] | 44.00 [28.00, 59.00] | 44.00 [28.00, 58.00] | | 47.00 [27.00, 59.00] | 46.00 [29.00, 58.00] | 0.0521 | 45.72 (20.06) | 45.14 (18.77) | 0.013 |
| | 44.00 [26.00, 59.00] | 44.00 [26.00, 36.00] | 0.0000 | 47.00 [27.00, 39.00] | 40.00 [29.00, 38.00] | 0.0321 | 45.72 (20.06) | 45.14 (16.77) | 0.030 |
| Age categories | 901 (17.3%) | 757 (14 69/) | 0.0068 | 1 206 (17 20/) | 029/12 E9/\ | 0.0097 | 2,107 (17.3%) | 1 605 (12 00/) | 0.094 |
| 12-17; n (%) | ` ' | 757 (14.6%) | | 1,206 (17.3%) | 938 (13.5%) | | | 1,695 (13.9%) | |
| 18-39; n (%) | 1,308 (25.2%) | 1,394 (26.8%) | -0.0031 | 1,566 (22.5%) | 1,677 (24.1%) | -0.0033 | 2,874 (23.6%) | 3,071 (25.3%) | -0.040 |
| 40 - 64; n (%) | 2,107 (40.5%) | 2,267 (43.6%) | -0.0048 | 3,281 (47.1%) | 3,660 (52.6%) | -0.0078 | 5,388 (44.3%) | 5,927 (48.8%) | -0.090 |
| >=65; n (%) | 882 (17.0%) | 780 (15.0%) | 0.0050 | 906 (13.0%) | 684 (9.8%) | 0.0095 | 1,788 (14.7%) | 1,464 (12.0%) | 0.079 |
| Geographic Region* | () | | | . === (== ===) | . === (==) | | | | |
| Northeast; n (%) | 715 (13.8%) | 748 (14.4%) | -0.0016 | 1,576 (22.6%) | 1,560 (22.4%) | 0.0004 | 2,291 (18.8%) | 2,308 (19.0%) | -0.005 |
| South; n (%) | 1,950 (37.5%) | 1,928 (37.1%) | 0.0007 | 2,066 (29.7%) | 2,040 (29.3%) | 0.0007 | 4,016 (33.0%) | 3,968 (32.6%) | 0.009 |
| Midwest; n (%) | 1,445 (27.8%) | 1,455 (28.0%) | -0.0004 | 2,220 (31.9%) | 2,261 (32.5%) | -0.0011 | 3,665 (30.1%) | 3,716 (30.6%) | -0.011 |
| West; n (%) | 1,088 (20.9%) | 1,067 (20.5%) | 0.0009 | 1,042 (15.0%) | 1,031 (14.8%) | 0.0005 | 2,130 (17.5%) | 2,098 (17.3%) | 0.005 |
| Unknown/Missing; n (%) | NA | NA | NA | 55 (0.8%) | 67 (1.0%) | -0.0021 | NA | NA | NA |
| Metropolitan Statistical Area* | | | | | | | | | |
| Urban; n (%) | NA | NA | NA | 5,712 (82.1%) | 5,672 (81.5%) | 0.0007 | NA | NA | NA |
| Rural; n (%) | NA | NA | NA | 108 (1.6%) | 104 (1.5%) | 0.0008 | NA | NA | NA |
| Unknown/Missing; n (%) | NA | NA | NA | 1,139 (16.4%) | 1,183 (17.0%) | -0.0015 | NA | NA | NA |
| General Health Related Measures | | | | | | | | | |
| Alcohol/Drug abuse or dependence ; n (%) | 12 (0.2%) | 26 (0.5%) | -0.0051 | 29 (0.4%) | 20 (0.3%) | 0.0017 | 041 (0.3%) | 046 (0.4%) | -0.017 |
| Obesity or Overweight; n (%)* | 319 (6.1%) | 293 (5.6%) | 0.0021 | 436 (6.3%) | 427 (6.1%) | 0.0008 | 755 (6.2%) | 720 (5.9%) | 0.013 |
| Obesity; n (%) | 258 (5.0%) | 251 (4.8%) | 0.0009 | 372 (5.3%) | 353 (5.1%) | 0.0009 | 630 (5.2%) | 604 (5.0%) | 0.009 |
| Overweight; n (%) | 63 (1.2%) | 50 (1.0%) | 0.0019 | 73 (1.0%) | 83 (1.2%) | -0.0019 | 136 (1.1%) | 133 (1.1%) | 0.000 |
| Cardiovascular Measures | | | | | | | | | |
| Hypertension; n (%)* | 1,300 (25.0%) | 1,268 (24.4%) | 0.0012 | 1,630 (23.4%) | 1,621 (23.3%) | 0.0002 | 2,930 (24.1%) | 2,889 (23.8%) | 0.007 |
| Hyperlipidemia; n (%)* | 1,109 (21.3%) | 1,050 (20.2%) | 0.0024 | 1,252 (18.0%) | 1,235 (17.7%) | 0.0007 | 2,361 (19.4%) | 2,285 (18.8%) | 0.015 |
| MI, angina, Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%)* | 176 (3.4%) | 159 (3.1%) | 0.0017 | 224 (3.2%) | 215 (3.1%) | 0.0006 | 400 (3.3%) | 374 (3.1%) | 0.011 |
| Old MI; n (%) | 17 (0.3%) | 15 (0.3%) | 0.0000 | 19 (0.3%) | 14 (0.2%) | 0.0020 | 036 (0.3%) | 029 (0.2%) | 0.020 |
| Acute MI; n (%) | 7 (0.1%) | 6 (0.1%) | 0.0000 | 11 (0.2%) | 4 (0.1%) | 0.0026 | 018 (0.1%) | 010 (0.1%) | 0.000 |
| Stable angina; n (%) | 25 (0.5%) | 31 (0.6%) | -0.0013 | 28 (0.4%) | 25 (0.4%) | 0.0000 | 053 (0.4%) | 056 (0.5%) | -0.015 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 159 (3.1%) | 134 (2.6%) | 0.0030 | 186 (2.7%) | 192 (2.8%) | -0.0006 | 345 (2.8%) | 326 (2.7%) | 0.006 |
| History of CABG or PTCA; n (%) | 29 (0.6%) | 26 (0.5%) | 0.0013 | 20 (0.3%) | 24 (0.3%) | 0.0000 | 049 (0.4%) | 050 (0.4%) | 0.000 |
| matery of Cabe of Frea, if (70) | 25 (0.070) | 20 (0.370) | 0.0013 | 20 (0.3/0) | 27 (0.370) | 0.0000 | 075 (0.470) | 030 (0.470) | 0.000 |

| _ | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%)* | 31 (0.6%) | 37 (0.7%) | -0.0012 | 58 (0.8%) | 58 (0.8%) | 0.0000 | 089 (0.7%) | 095 (0.8%) | -0.012 |
| Stroke (Ischemic or hemorrhagic); n (%) | 17 (0.3%) | 20 (0.4%) | -0.0017 | 23 (0.3%) | 35 (0.5%) | -0.0032 | 040 (0.3%) | 055 (0.5%) | -0.032 |
| TIA; n (%) | 11 (0.2%) | 14 (0.3%) | -0.0020 | 32 (0.5%) | 26 (0.4%) | 0.0015 | 043 (0.4%) | 040 (0.3%) | 0.017 |
| Late effects of cerebrovascular disease; n (%) | 8 (0.2%) | 9 (0.2%) | 0.0000 | 12 (0.2%) | 13 (0.2%) | 0.0000 | 020 (0.2%) | 022 (0.2%) | 0.000 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%)* | 200 (3.8%) | 191 (3.7%) | 0.0005 | 312 (4.5%) | 312 (4.5%) | 0.0000 | 512 (4.2%) | 503 (4.1%) | 0.005 |
| Atrial fibrillation; n (%) | 96 (1.8%) | 89 (1.7%) | 0.0008 | 158 (2.3%) | 123 (1.8%) | 0.0035 | 254 (2.1%) | 212 (1.7%) | 0.029 |
| Other cardiac dysrhythmia; n (%) | 136 (2.6%) | 138 (2.7%) | -0.0006 | 209 (3.0%) | 242 (3.5%) | -0.0028 | 345 (2.8%) | 380 (3.1%) | -0.018 |
| Diabetes Related Measures | | | | | | | | | |
| Diabetes with or w/o complications; n (%)* | 411 (7.9%) | 354 (6.8%) | 0.0041 | 496 (7.1%) | 503 (7.2%) | -0.0004 | 907 (7.5%) | 857 (7.0%) | 0.019 |
| Diabetes mellitus without mention of complications; n (%) | 395 (7.6%) | 329 (6.3%) | 0.0049 | 463 (6.7%) | 481 (6.9%) | -0.0008 | 858 (7.1%) | 810 (6.7%) | 0.016 |
| Diabetes with specified complications; n (%) | 73 (1.4%) | 57 (1.1%) | 0.0027 | 83 (1.2%) | 66 (0.9%) | 0.0029 | 156 (1.3%) | 123 (1.0%) | 0.028 |
| Diabetes with unspecified complications; n (%) | 16 (0.3%) | 13 (0.3%) | 0.0000 | 17 (0.2%) | 14 (0.2%) | 0.0000 | 033 (0.3%) | 027 (0.2%) | 0.020 |
| GI Conditions | | | | | | | | | |
| GERD; n (%)* | 492 (9.5%) | 467 (9.0%) | 0.0016 | 591 (8.5%) | 611 (8.8%) | -0.0010 | 1,083 (8.9%) | 1,078 (8.9%) | 0.000 |
| Upper GI (Diseases of esophagus, stomach and duodenum including GERD); n (%) | 611 (11.8%) | 597 (11.5%) | 0.0009 | 763 (11.0%) | 783 (11.3%) | -0.0009 | 1,374 (11.3%) | 1,380 (11.4%) | -0.003 |
| GI bleeding; n (%)* | 71 (1.4%) | 63 (1.2%) | 0.0018 | 77 (1.1%) | 94 (1.4%) | -0.0027 | 148 (1.2%) | 157 (1.3%) | -0.009 |
| Non-infective enteritis and colitis; n (%) | 153 (2.9%) | 164 (3.2%) | -0.0017 | 229 (3.3%) | 215 (3.1%) | 0.0011 | 382 (3.1%) | 379 (3.1%) | 0.000 |
| Intraoperative and postprocedural complications and disorders of digestive system; n (%) | 75 (1.4%) | 55 (1.1%) | 0.0027 | 71 (1.0%) | 70 (1.0%) | 0.0000 | 146 (1.2%) | 125 (1.0%) | 0.019 |
| - | 42 (0.00/) | 40 (0.00() | 0.0000 | F.C. (O. 90/.) | F7 (0.00/) | 0.0000 | 000 (0.00/) | 007 (0.0%) | 0.000 |
| Disorders of gallbladder, biliary tract and pancreas; n (%)* | 42 (0.8%) | 40 (0.8%) | 0.0000 | 56 (0.8%) | 57 (0.8%) | 0.0000 | 098 (0.8%) | 097 (0.8%) | 0.000 |
| Rheumatic Conditions | | | | | | | | | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n<br>(%)* | 59 (1.1%) | 52 (1.0%) | 0.0010 | 100 (1.4%) | 108 (1.6%) | -0.0016 | 159 (1.3%) | 160 (1.3%) | 0.000 |
| Osteoarthrosis; n (%)* | 366 (7.0%) | 347 (6.7%) | 0.0011 | 525 (7.5%) | 498 (7.2%) | 0.0011 | 891 (7.3%) | 845 (7.0%) | 0.012 |
| Other rheumatic disorders (including gout); n (%)* | 1,007 (19.4%) | 989 (19.0%) | 0.0009 | 1,405 (20.2%) | 1,420 (20.4%) | -0.0004 | 2,412 (19.8%) | 2,409 (19.8%) | 0.000 |
| Gout and other crystal arthropathies; n (%) | 35 (0.7%) | 41 (0.8%) | -0.0012 | 35 (0.5%) | 55 (0.8%) | -0.0037 | 070 (0.6%) | 096 (0.8%) | -0.024 |
| Other rheumatic disorders; n (%) | 988 (19.0%) | 960 (18.5%) | 0.0012 | 1,382 (19.9%) | 1,381 (19.8%) | 0.0002 | 2,370 (19.5%) | 2,341 (19.3%) | 0.005 |
| Neuro Conditions* | | | | | | | | | |
| Alzheimer and other Dementia Disease ; n (%) | 35 (0.7%) | 31 (0.6%) | 0.0012 | 30 (0.4%) | 37 (0.5%) | -0.0015 | 065 (0.5%) | 068 (0.6%) | -0.014 |
| Seizure disorders (epilepsy); n (%) | 26 (0.5%) | 28 (0.5%) | 0.0000 | 40 (0.6%) | 41 (0.6%) | 0.0000 | 066 (0.5%) | 069 (0.6%) | -0.014 |
| Delirium/Psychosis; n (%) | 44 (0.8%) | 43 (0.8%) | 0.0000 | 43 (0.6%) | 46 (0.7%) | -0.0012 | 087 (0.7%) | 089 (0.7%) | 0.000 |
| Other Conditions | | | | | | | | | |
| Hypothyroidism; n (%)* | 484 (9.3%) | 484 (9.3%) | 0.0000 | 531 (7.6%) | 512 (7.4%) | 0.0007 | 1,015 (8.3%) | 996 (8.2%) | 0.004 |
| Chronic kidney disease stages I-III; n (%)* | 100 (1.9%) | 101 (1.9%) | 0.0000 | 59 (0.8%) | 60 (0.9%) | -0.0011 | 159 (1.3%) | 161 (1.3%) | 0.000 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 31 (0.6%) | 25 (0.5%) | 0.0013 | 17 (0.2%) | 16 (0.2%) | 0.0000 | 048 (0.4%) | 041 (0.3%) | 0.017 |
| COPD; n (%)* | 261 (5.0%) | 258 (5.0%) | 0.0000 | 352 (5.1%) | 347 (5.0%) | 0.0004 | 613 (5.0%) | 605 (5.0%) | 0.000 |
| Obstructive sleep apnea; n (%)* | 274 (5.3%) | 263 (5.1%) | 0.0009 | 372 (5.3%) | 378 (5.4%) | -0.0004 | 646 (5.3%) | 641 (5.3%) | 0.000 |
| Syncope; n (%) | 62 (1.2%) | 50 (1.0%) | 0.0019 | 72 (1.0%) | 86 (1.2%) | -0.0019 | 134 (1.1%) | 136 (1.1%) | 0.000 |
| Falls; n (%) | 58 (1.1%) | 42 (0.8%) | 0.0031 | 39 (0.6%) | 30 (0.4%) | 0.0028 | 097 (0.8%) | 072 (0.6%) | 0.024 |
| VTE; n (%)* | 32 (0.6%) | 36 (0.7%) | -0.0012 | 57 (0.8%) | 59 (0.8%) | 0.0000 | 089 (0.7%) | 095 (0.8%) | -0.012 |
| Combined comorbidity score, 365 days* | | | | | | | | | |
| mean (sd) | 1.17 (0.96) | 1.15 (0.97) | 0.0207 | 1.15 (0.89) | 1.13 (0.86) | 0.0229 | 1.16 (0.92) | 1.14 (0.91) | 0.022 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 (0.92) | 1.00 (0.91) | 0.000 |
| Frailty Score: Empirical Version 365 days as Categories* | | | | | | | | | |
| < 0.1 non frail; n (%) | 3,483 (67.0%) | 3,450 (66.4%) | 0.0007 | 4,163 (59.8%) | 4,169 (59.9%) | -0.0001 | 7,646 (62.9%) | 7,619 (62.7%) | 0.004 |
| 0.1 -< 0.2 prefrail; n (%) | 1,118 (21.5%) | 1,168 (22.5%) | -0.0021 | 1,741 (25.0%) | 1,748 (25.1%) | -0.0002 | 2,859 (23.5%) | 2,916 (24.0%) | -0.012 |
| > 0.2 frail; n (%) | 597 (11.5%) | 580 (11.2%) | 0.0009 | 1,055 (15.2%) | 1,042 (15.0%) | 0.0005 | 1,652 (13.6%) | 1,622 (13.3%) | 0.009 |
| Medication Use | | | | | | | | | |
| Use of oral corticosteroids; n (%)* | 2,474 (47.6%) | 2,528 (48.6%) | -0.0014 | 6,612 (95.0%) | 6,635 (95.3%) | -0.0003 | 9,086 (74.7%) | 9,163 (75.4%) | -0.01 |
| Use of antidepressants; n (%)* | 981 (18.9%) | 984 (18.9%) | 0.0000 | 1,520 (21.8%) | 1,525 (21.9%) | -0.0002 | 2,501 (20.6%) | 2,509 (20.6%) | 0.000 |
| Use of anticonvulsants; n (%)* | 297 (5.7%) | 284 (5.5%) | 0.0008 | 509 (7.3%) | 487 (7.0%) | 0.0011 | 806 (6.6%) | 771 (6.3%) | 0.012 |
| Use of beta blocker OR calcium channel blocker; n (%)* | 505 (9.7%) | 474 (9.1%) | 0.0020 | 751 (10.8%) | 732 (10.5%) | 0.0009 | 1,256 (10.3%) | 1,206 (9.9%) | 0.013 |
| Use of PPIs; n (%)* | 744 (14.3%) | 734 (14.1%) | 0.0005 | 1,413 (20.3%) | 1,430 (20.5%) | -0.0004 | 2,157 (17.7%) | 2,164 (17.8%) | -0.003 |

| Use of opioids; n (%)* | 808 (15.5%) | 781 (15.0%) | 0.0013 | 1,307 (18.8%) | 1,308 (18.8%) | 0.0000 | 2,115 (17.4%) | 2,089 (17.2%) | 0.005 |
|---|---|---|---|---|---|---|---|---|---|
| Use of antipsychotics; n (%)* | 73 (1.4%) | 73 (1.4%) | 0.0000 | 101 (1.5%) | 99 (1.4%) | 0.0008 | 174 (1.4%) | 172 (1.4%) | 0.000 |
| Use of anxiolytics/hypnotics; n (%)* | 289 (5.6%) | 285 (5.5%) | 0.0004 | 457 (6.6%) | 489 (7.0%) | -0.0015 | 746 (6.1%) | 774 (6.4%) | -0.012 |
| Use of dementia meds; n (%)* | 23 (0.4%) | 23 (0.4%) | 0.0004 | 21 (0.3%) | 23 (0.3%) | 0.0000 | 044 (0.4%) | 046 (0.4%) | 0.000 |
| Use of antiparkinsonian meds; n (%)* | 53 (1.0%) | 51 (1.0%) | 0.0000 | 98 (1.4%) | 103 (1.5%) | -0.0008 | 151 (1.2%) | 154 (1.3%) | -0.009 |
| Use of Benzodiazepine; n (%)* | 467 (9.0%) | 454 (8.7%) | 0.0010 | 822 (11.8%) | 839 (12.1%) | -0.0009 | 1,289 (10.6%) | 1,293 (10.6%) | 0.000 |
| All antidiabetic medications; n (%)* | 328 (6.3%) | 286 (5.5%) | 0.0010 | 474 (6.8%) | 491 (7.1%) | -0.0003 | 802 (6.6%) | 777 (6.4%) | 0.008 |
| ACEI/ARB; n (%)8 | 875 (16.8%) | 865 (16.6%) | 0.0033 | 1,316 (18.9%) | 1,334 (19.2%) | -0.0011 | 2,191 (18.0%) | 2,199 (18.1%) | -0.003 |
| Use of Anticoagulants; n (%)* | 104 (2.0%) | 91 (1.8%) | 0.0005 | 154 (2.2%) | 150 (2.2%) | 0.0000 | 258 (2.1%) | 241 (2.0%) | 0.003 |
| Use of Amiodarone; n (%) | 9 (0.2%) | 10 (0.2%) | 0.0000 | 16 (0.2%) | 9 (0.1%) | 0.0026 | 025 (0.2%) | 019 (0.2%) | 0.000 |
| Digoxin; n (%) | 22 (0.4%) | 17 (0.3%) | 0.0007 | 41 (0.6%) | 30 (0.4%) | 0.0028 | 063 (0.5%) | 047 (0.4%) | 0.015 |
| Use of Diuretics; n (%)* | 705 (13.6%) | 689 (13.3%) | 0.0017 | 1,104 (15.9%) | 1,108 (15.9%) | 0.0028 | 1,809 (14.9%) | 1,797 (14.8%) | 0.013 |
| Use of Aspirin; n (%) | 16 (0.3%) | 17 (0.3%) | 0.0000 | 25 (0.4%) | 27 (0.4%) | 0.0000 | 041 (0.3%) | 044 (0.4%) | -0.017 |
| NSAIDs (NOT including aspirin); n (%) | 463 (8.9%) | 523 (10.1%) | -0.0039 | 811 (11.7%) | 929 (13.3%) | -0.0045 | 1,274 (10.5%) | 1,452 (11.9%) | -0.044 |
| HRT (Use of estrogens, progestins, androgens); n (%)* | 716 (13.8%) | 735 (14.1%) | -0.0008 | 1,088 (15.6%) | 1,111 (16.0%) | -0.0010 | 1,804 (14.8%) | 1,846 (15.2%) | -0.011 |
| Use of Statins; n (%)* | 909 (17.5%) | 870 (16.7%) | 0.0019 | 1,203 (17.3%) | 1,188 (17.1%) | 0.0005 | 2,112 (17.4%) | 2,058 (16.9%) | 0.011 |
| Healthcare Utilization Measures | 303 (17.3%) | 070 (10.770) | 0.0013 | 1,203 (17.370) | 1,100 (17.170) | 0.0003 | 2,112 (17.470) | 2,030 (10.370) | 0.015 |
| Use of any drugs claims* | | | | | | | | | |
| mean (sd) | 22.17 (17.48) | 22.00 (16.75) | 0.0099 | 24.51 (16.99) | 24.60 (17.10) | -0.0053 | 23.51 (17.20) | 23.49 (16.95) | 0.001 |
| median [IQR] | 18.00 [10.00, 29.00] | 18.00 [10.00, 29.00] | | 20.00 [12.00, 32.00] | 21.00 [12.00, 32.00] | -0.0587 | 19.14 (17.20) | 19.72 (16.95) | -0.034 |
| Number of office visits* | 10.00 [10.00, 25.00] | 10.00 [10.00, 25.00] | 0.0000 | 20.00 [12.00, 32.00] | 21.00 [12.00, 32.00] | 0.0307 | 15.14 (17.20) | 15.72 (10.55) | 0.054 |
| mean (sd) | 10.07 (8.28) | 10.04 (8.68) | 0.0035 | 11.05 (8.13) | 11.08 (7.78) | -0.0038 | 10.63 (8.19) | 10.64 (8.18) | -0.001 |
| median [IQR] | 8.00 [5.00, 13.00] | 8.00 [5.00, 12.25] | 0.0000 | 9.00 [6.00, 14.00] | 9.00 [6.00, 14.00] | 0.0000 | 8.57 (8.19) | 8.57 (8.18) | 0.000 |
| Number of ED visits* | 0.00 [5.00, 15.00] | 0.00 [5.00, 12.25] | 0.0000 | 3.00 [0.00, 14.00] | 5.00 [0.00, 14.00] | 0.0000 | 0.57 (0.15) | 0.57 (0.10) | 0.000 |
| mean (sd) | 0.33 (0.77) | 0.32 (0.76) | 0.0131 | 0.52 (1.15) | 0.52 (1.07) | 0.0000 | 0.44 (1.01) | 0.43 (0.95) | 0.010 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (1.01) | 0.00 (0.95) | 0.000 |
| Number of hospitalizations* | 0.00 [0.00) 0.00] | 0.00 [0.00) 0.00] | 0.0000 | 0.00 [0.00) 2.00] | 0.00 [0.00, 2.00] | 0.0000 | 0.00 (1.01) | 0.00 (0.55) | 0.000 |
| mean (sd) | 0.03 (0.20) | 0.03 (0.25) | 0.0000 | 0.16 (1.29) | 0.14 (1.09) | 0.0167 | 0.10 (0.98) | 0.09 (0.84) | 0.011 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.98) | 0.00 (0.84) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%)* | 14 (0.3%) | 8 (0.2%) | 0.0020 | 38 (0.5%) | 40 (0.6%) | -0.0013 | 052 (0.4%) | 048 (0.4%) | 0.000 |
| Old hospitalizations (-365 to -31 days); n (%)* | 295 (5.7%) | 303 (5.8%) | -0.0004 | 468 (6.7%) | 482 (6.9%) | -0.0008 | 763 (6.3%) | 785 (6.5%) | -0.008 |
| Number of Pulmonologist/Allergist visits* | | (5.5.5) | | | | | ( , . , | ( , | |
| mean (sd) | 0.02 (0.26) | 0.02 (0.27) | 0.0000 | 1.38 (3.64) | 1.39 (3.52) | -0.0028 | 0.80 (2.76) | 0.80 (2.67) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (2.76) | 0.00 (2.67) | 0.000 |
| Pulmonologist /allergist on CED; n (%)* | 3 (0.1%) | 2 (0.0%) | 0.0045 | 456 (6.6%) | 466 (6.7%) | -0.0004 | 459 (3.8%) | 468 (3.8%) | 0.000 |
| Number of hospital days* | | | | | | | | | |
| mean (sd) | 0.21 (2.95) | 0.19 (2.73) | 0.0070 | 0.16 (1.29) | 0.14 (1.09) | 0.0167 | 0.18 (2.16) | 0.16 (1.97) | 0.010 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (2.16) | 0.00 (1.97) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood chemistry | | | 0.0004 | | | 0.0004 | | | 0.044 |
| test; n (%)* | 1,406 (27.0%) | 1,348 (25.9%) | 0.0021 | 1,693 (24.3%) | 1,679 (24.1%) | 0.0004 | 3,099 (25.5%) | 3,027 (24.9%) | 0.014 |
| Number of HbA1C test ordered* | | | | | | | | | |
| mean (sd) | 0.33 (0.88) | 0.29 (0.80) | 0.0476 | 0.29 (0.78) | 0.29 (0.78) | 0.0000 | 0.31 (0.82) | 0.29 (0.79) | 0.025 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.82) | 0.00 (0.79) | 0.000 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; | 162 (3.1%) | 159 (3.1%) | 0.0000 | 236 (3.4%) | 244 (3.5%) | -0.0005 | 398 (3.3%) | 403 (3.3%) | 0.000 |
| n (%)* | 102 (5.1%) | 139 (3.1%) | 0.0000 | 250 (5.4%) | 244 (3.5%) | -0.0003 | 390 (3.3%) | 403 (3.3%) | 0.000 |
| Number of Mammograms (Breast cancer screening); n (%)* | 687 (13.2%) | 669 (12.9%) | 0.0008 | 918 (13.2%) | 918 (13.2%) | 0.0000 | 1,605 (13.2%) | 1,587 (13.1%) | 0.003 |
| Number of Pap smear (Cervical cancer screening); n (%)* | 690 (13.3%) | 707 (13.6%) | -0.0008 | 961 (13.8%) | 954 (13.7%) | 0.0003 | 1,651 (13.6%) | 1,661 (13.7%) | -0.003 |
| Flu vaccine; n (%)* | 973 (18.7%) | 982 (18.9%) | -0.0005 | 1,201 (17.3%) | 1,155 (16.6%) | 0.0017 | 2,174 (17.9%) | 2,137 (17.6%) | 0.008 |
| Pneumococcal vaccine; n (%)* | 307 (5.9%) | 306 (5.9%) | 0.0000 | 443 (6.4%) | 448 (6.4%) | 0.0000 | 750 (6.2%) | 754 (6.2%) | 0.000 |
| Copay for pharmacy cost (charges in U.S. \$)* | | | | | | | | | |
| mean (sd) | 35.89 (33.14) | 36.20 (29.55) | -0.0099 | 25.00 (23.64) | 24.90 (23.97) | 0.0042 | 29.66 (28.10) | 29.73 (26.50) | -0.003 |
| median [IQR] | 29.37 [16.66, 46.02] | 31.05 [18.46, 47.50] | -0.0535 | 21.00 [9.54, 34.19] | 20.80 [10.00, 34.36] | 0.0084 | 24.58 (28.10) | 25.18 (26.50) | -0.022 |
| Business Type* | | | | | | | | | |
| Commercial; n (%) | 4,456 (85.7%) | 4,494 (86.5%) | -0.0009 | NA | NA | NA | NA | NA | NA |

| Medicare; n (%) | 742 (14.3%) | 704 (13.5%) | 0.0021 | NA | NA | NA | NA | NA | NA |
|---|---|---|---|---|---|---|---|---|---|
| Insurance Plan Type* | | | | | | | | | |
| Comprehensive; n (%) | NA | NA | NA | 547 (7.9%) | 554 (8.0%) | -0.0004 | NA | NA | NA |
| HMO; n (%) | NA | NA | NA | 902 (13.0%) | 896 (12.9%) | 0.0003 | NA | NA | NA |
| PPO; n (%) | NA | NA | NA | 4,037 (58.0%) | 4,052 (58.2%) | -0.0003 | NA | NA | NA |
| Others; n (%) | NA | NA | NA | 1,473 (21.2%) | 1,457 (20.9%) | 0.0007 | NA | NA | NA |
| SABA; n (%)* | 2,756 (53.0%) | 2,770 (53.3%) | -0.0004 | 4,454 (64.0%) | 4,477 (64.3%) | -0.0004 | 7,210 (59.3%) | 7,247 (59.6%) | -0.006 |
| SAMA; n (%)* | 79 (1.5%) | 66 (1.3%) | 0.0017 | 182 (2.6%) | 187 (2.7%) | -0.0006 | 261 (2.1%) | 253 (2.1%) | 0.000 |
| SABA/SAMA; n (%)* | 101 (1.9%) | 100 (1.9%) | 0.0000 | 255 (3.7%) | 265 (3.8%) | -0.0005 | 356 (2.9%) | 365 (3.0%) | -0.006 |
| ICS without budesonide; n (%)* | 1,600 (30.8%) | 1,649 (31.7%) | -0.0016 | 2,596 (37.3%) | 2,705 (38.9%) | -0.0026 | 4,196 (34.5%) | 4,354 (35.8%) | -0.027 |
| LABA; n (%)* | 209 (4.0%) | 191 (3.7%) | 0.0015 | 340 (4.9%) | 349 (5.0%) | -0.0004 | 549 (4.5%) | 540 (4.4%) | 0.005 |
| LAMA; n (%)* | 111 (2.1%) | 115 (2.2%) | -0.0007 | 228 (3.3%) | 243 (3.5%) | -0.0011 | 339 (2.8%) | 358 (2.9%) | -0.006 |
| ICS/LABA (without budesonide-formoterol); n (%)* | 546 (10.5%) | 568 (10.9%) | -0.0012 | 813 (11.7%) | 857 (12.3%) | -0.0017 | 1,359 (11.2%) | 1,425 (11.7%) | -0.016 |
| Blood eosinophilia test ; n (%)* | 15 (0.3%) | 16 (0.3%) | 0.0000 | 13 (0.2%) | 15 (0.2%) | 0.0000 | 028 (0.2%) | 031 (0.3%) | -0.020 |
| Serum immunoglobulin E (IgE) level test; n (%)* | 62 (1.2%) | 72 (1.4%) | -0.0018 | 119 (1.7%) | 119 (1.7%) | 0.0000 | 181 (1.5%) | 191 (1.6%) | -0.008 |
| H2 blocker; n (%)* | 56 (1.1%) | 60 (1.2%) | -0.0009 | 213 (3.1%) | 193 (2.8%) | 0.0017 | 269 (2.2%) | 253 (2.1%) | 0.007 |
| Oxygen codes; n (%)* | 14 (0.3%) | 7 (0.1%) | 0.0045 | 32 (0.5%) | 29 (0.4%) | 0.0015 | 046 (0.4%) | 036 (0.3%) | 0.017 |
| Respiratory arrest/dependence on oxygen; n (%)* | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 001 (0.0%) | 000 (0.0%) | #DIV/0! |

<sup>\*</sup>Included in the 1:1 PS matching model